CLINICAL TRIAL: NCT00546871
Title: Tolerability and Pharmacokinetic Comparison of Immune Globulin Intravenous (Human) 10% (IGIV, 10%) Administered Intravenously or Subcutaneously in Subjects With Primary Immunodeficiency Diseases
Brief Title: Comparison of Intravenous and Subcutaneous Administration of IGIV, 10% in Primary Immunodeficiency (PID) Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160601
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human), 10% — Intravenous administration in Study Part 1, subcutaneous administration in Study Parts 2 and 3

SUMMARY:
The purpose of this study is to evaluate the tolerability of IGIV, 10% given subcutaneously and the pharmacokinetics of immunoglobulin G (IgG) following subcutaneous (SC) treatment with IGIV, 10% in subjects with primary immunodeficiency (PID) disorders.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from either the subject or the subject's legally acceptable representative prior to any study-related procedures and study product administration
* Diagnosis of a PID disorder as defined by World Health Organization criteria (IUIS Scientific Committee, Primary immunodeficiency diseases. Report of an IUIS Scientific Committee. Clin Exp Immunol. 1999) for which the subject has been receiving a regular regimen of IV immunoglobulin infusions every 21 ± 3 days or 28 ± 3 days or a regular SC immunoglobulin treatment at 1 to 2 week intervals over a period of at least 3 months pre-study at a dose of 300-800 mg/kg BW/4 weeks
* Subjects are aged 2 years or older
* Subjects have a serum trough level of IgG > 4.5 g/L at the last documented determination
* A negative serum pregnancy test for any female subject who is of childbearing potential
* Female subjects of childbearing potential agree to practice birth control measures for the duration of the study

Exclusion Criteria:

* Subjects positive at enrollment for one or more of the following: Hepatitis B surface antigen (HBsAg), PCR for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1
* Subjects with levels of alanine amino transferase (ALT) or aspartate amino transferase (AST) > 2.5 times the upper limit of normal for the testing laboratory
* Subjects with neutropenia (defined as an absolute neutrophil count [ANC] <= 500/mm3)
* Subjects with serum creatinine levels greater than 1.5 times the upper limit of normal for age and gender
* Subjects with a malignancy other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Subjects with a history of thrombotic episodes (deep vein thrombosis, myocardial infarction, cerebrovascular accident)
* Subjects with abnormal protein loss (protein losing enteropathy, nephritic syndrome, severe lung disease)
* Subjects with anemia that would preclude phlebotomy for laboratory studies
* Subjects who received any blood or blood product other than an IGIV, SC immunoglobulin, immune serum globulin (ISG) preparation, or albumin within the 6 months prior to study enrollment
* Subjects with an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IGIV, SC immunoglobulin and/or ISG infusions
* Subjects with IgA deficiency and known anti IgA antibodies
* Subjects receiving antibiotic therapy for the treatment of infection within 7 days prior to enrollment
* Subjects participating in another clinical study involving an investigational product or device within 28 days prior to study enrollment
* Subjects with bleeding disorders or who are on anti-coagulation therapy

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-10-03 (Actual); Primary Completion 2009-07-01 (Actual); Study Completion 2009-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (9):
  - Los Angeles, California
  - Centennial, Colorado
  - North Palm Beach, Florida
  - Atlanta, Georgia
  - Durham, North Carolina
  - Cleveland, Ohio
  - Dallas, Texas
  - Galveston, Texas
  - Milwaukee, Wisconsin

REFERENCES:
- [Background] Neu AM, Warady BA, Furth SL, Lederman HM, Fivush BA. Antibody levels to diphtheria, tetanus, and rubella in infants vaccinated while on PD: a Study of the Pediatric Peritoneal Dialysis Study Consortium. Adv Perit Dial. 1997;13:297-9. PMID 9440877
- [Result] Leibl H, Engl W, Melamed I, Stein M, Wasserman RL, Berger M, Schiff RI. IGIV-10% Infused Intravenously And Subcutaneously To Subjects With Primary Immunodeficiency Diseases - Comparison Of Pharmacokinetic Properties. Poster presentation at AAAAI 2009.
- [Result] Schiff RI, Leibl H, Engl W. Pharmacokinetic properties of Gammagard Liquid 10% (KIOVIG) administered intravenously and subcutaneously to patients with primary immunodeficiency diseases. Clin Exp Immunol. 154 (Suppl. 1):132, 2008
- [Result] Wasserman RL, Melamed I, Kobrynski L, Strausbaugh SD, Stein MR, Sharkhawy M, Engl W, Leibl H, Sobolevsky L, Gelmont D, Schiff RI, Grossman WJ. Efficacy, safety, and pharmacokinetics of a 10% liquid immune globulin preparation (GAMMAGARD LIQUID, 10%) administered subcutaneously in subjects with primary immunodeficiency disease. J Clin Immunol. 2011 Jun;31(3):323-31. doi: 10.1007/s10875-011-9512-z. Epub 2011 Mar 22. PMID 21424824
- [Derived] Wasserman RL, Gupta S, Stein M, Rabbat CJ, Engl W, Leibl H, Yel L. Infection rates and tolerability of three different immunoglobulin administration modalities in patients with primary immunodeficiency diseases. Immunotherapy. 2022 Mar;14(4):215-224. doi: 10.2217/imt-2021-0256. Epub 2021 Dec 21. PMID 34931880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the United States at 9 study sites.
Pre-assignment Details: 53 participants who enrolled were screened. Of these, 4 withdrew before treatment (1 death, 1 screen failure, 2 requested withdrawal)
Groups:
- 2 to <12 Years; 12 Years and Older: Part 1: IV infusions of IGIV, 10% (every 3 or 4 weeks) for 12 weeks at dose/schedule prior to study (300 - 1,000 mg/kg/4 weeks). Pharmacokinetic (PK) done on ≥12 years after 3rd or 4th infusion Part 2: Weekly subcutaneous (SC) IGIV, 10% at 130% of weekly equivalent dose in Part 1 for ≥12 weeks, until 15 subjects ≥ 12years completed PK assessment. PK determined "Adjusted Dose" in Part 3a Part 3a: 6 weeks SC IGIV Adjusted Dose. Trough levels determined at Week 5 to see if increase in trough levels was not within 15% of expected increase, then dose was individually adapted Part 3b: Participants received weekly SC infusions for 12 weeks. Dose administered was determined as follows: -If trough levels within 15% of expected over trough level determined in Part 1, dosing remained same as Part 3a -If trough levels not within 15% of expected over trough level in Part 1, participants received Individually Adapted Dose Study Extension: Participants were offered to enter into Extension
Period: Part 1 - IV Infusions of IGIV, PK
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 14 | 35
Completed | 13 | 35
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Part 2 - Subcutaneous (SC) IGIV, PK
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 13 | 35
Completed | 12 | 32
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Family Emergency | 0 | 1
Period: Part 3a- SC IGIV Adjusted Dose, PK Based
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 12 | 32
Completed | 12 | 32
Not Completed | 0 | 0
Period: Part 3b - SC IGIV 12 Weeks
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 12 | 32
Completed | 12 | 32
Not Completed | 0 | 0
Period: Study Extension Period
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 10 (2 withdrawn after Part 3b) | 26 (6 withdrawn after Part 3b)
Completed | 9 | 25
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treated Participants
Number analyzed (Participants) | 49
Age, Customized [Count of Participants; unit: Participants]
  2 to <12 years | 14
  ≥ 12 years | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Area Under the Concentration Curve (AUC 0-τ)/Week Following IV Administration to SC Administration of IGIV, 10% at an Adjusted/Individual Adapted Dose (Part 3b), Expressed as a Percentage
Description: Expressed as (AUC_SC/AUC_IV) * 100
Time Frame: Week 12 (IV) and week 32 or 33 (SC)
Population: Participants, ≥12 years, with PK data in terms of AUC[0-τ]/week following IV administration and SC administration of IGIV, 10% at an adjusted/individually adapted dose in Study Part 3b
Measure: Number (90% Confidence Interval); unit: percent
Groups:
- Participants ≥12 Years Old With PK Data Part 1 and Part 3b: IV infusions of IGIV, 10% (every 3 or 4 weeks, ± 2 days) for 12 weeks at dose and schedule they were on prior to study (300 to 1,000 mg/kg/4 weeks). SC dosing for Study Part 3b was determined by: From Study Part 2, PK: Participants received weekly (± 1 day) SC IGIV at a dose of 130% of weekly equivalent of IV dose. First 15 participants ≥12 years to complete PK were used to determine the "Adjusted Dose". Study Part 3a, Adjusted Dose: Participants treated SC for 6 weeks using Adjusted Dose. If Adjusted Dose did not achieve expected trough levels, dose was adjusted to an "Individually Adapted Dose" to ensure sufficient trough levels. Study Part 3b: Participants received weekly SC infusions for 12 weeks. Dose administered was either: 1. The Adjusted Dose 2. Individually Adapted Dose
Arm/Group | Participants ≥12 Years Old With PK Data Part 1 and Part 3b
Number analyzed (Participants) | 29
percent | 95.2 [92.3 to 98.2]

2. Primary Outcome: Bioavailability (Trough Levels) of IgG After Administration of IGIV, 10%, in Participants Aged 2 to <12 Years.
Description: Administration of IGIV, 10%: - Part 1 = IV administration (IV) - Parts 2, 3a, 3b = SC administration (SC)
Time Frame: Baseline; at each 3 or 4-week study visit in Study Part 1; at Visits 1, 5, and 9 in Study Part 2; at Visits 1, and 5 in Study Part 3a; at Visits 1, 5, and 9 in Study Part 3b; and at the end-of-study evaluation
Population: Full safety data set (all participants, aged 2 to <12 years who received any study drug)
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | Participants Aged 2 to <12 Years
Number analyzed (Participants) | 14
g/L
  Part 1 (IV), Screening visit (n=14) | 11.400 [9.640 to 16.800]
  Part 1 (IV), 3 week Interval, Visit 1 (n=5) | 10.100 [NA to NA] — Evaluable sample size was too small
  Part 1 (IV), 3 week Interval, Visit 2 (n=4) | 11.500 [NA to NA] — Evaluable sample size was too small
  Part 1 (IV), 3 week Interval, Visit 3 (n=5) | 10.600 [NA to NA] — Evaluable sample size was too small
  Part 1 (IV), 3 week Interval, Visit 4 (n=5) | 10.100 [NA to NA] — Evaluable sample size was too small
  Part 1 (IV), 3 week Interval, Visit 5 (n=5) | 10.800 [NA to NA] — Evaluable sample size was too small
  Part 1 (IV), 4 week Interval, Visit 1 (n=7) | 9.640 [7.240 to 17.400]
  Part 1 (IV), 4 week Interval, Visit 2 (n=9) | 10.000 [7.230 to 12.400]
  Part 1 (IV), 4 week Interval, Visit 3 (n=7) | 9.080 [6.340 to 18.500]
  Part 1 (IV), 4 week Interval, Visit 4 (n=8) | 10.500 [7.420 to 17.800]
  Part 2 (SC), Visit 1 (n=12) | 13.650 [12.300 to 16.700]
  Part 2 (SC), Visit 5 (n=12) | 12.800 [11.200 to 16.500]
  Part 2 (SC), Visit 9 (n=12) | 13.600 [10.100 to 17.100]
  Part 3a (SC), Visit 1 (n=11) | 11.200 [10.300 to 19.100]
  Part 3a (SC), Visit 5 (n=11) | 12.200 [11.500 to 20.000]
  Part 3b (SC), Visit 1 (n=12) | 11.500 [9.170 to 15.800]
  Part 3b (SC), Visit 5 (n=12) | 12.600 [10.200 to 15.200]
  Part 3b (SC), Visit 9 (n=12) | 12.800 [10.300 to 15.900]
  End of Study (n=13) | 12.300 [8.570 to 18.000]

3. Secondary Outcome: Study Part 1 (IV): Maximum Plasma Concentration (C-max)
Description: Maximal immune globulin concentration after infusion
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #3 starts) up to 28 days (+/-2 days) post-infusion.
Population: Participants for whom the following PK measurements are available: 1. pre-infusion and the 30-minute-post-infusion measurements 2. ≥3 measurements for Days 1, 4, 9, 14, and 21 and/or 28 3. for the 3-week treatment schedule: Day 14 and/or the Day 21 measurement(s); for the 4-week treatment schedule: Day 21 and/or the Day 28 measurement(s)
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
g/L | 22.7 [21.0 to 25.0]

4. Secondary Outcome: Study Part 1 (IV): Minimum Plasma Concentration (C-min)
Description: Minimal immune globulin concentration after infusion
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
g/L | 10.1 [9.4 to 12.4]

5. Secondary Outcome: Study Part 1 (IV): Weight-adjusted Clearance
Description: Computed as weight-adjusted dose divided by total AUC
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: mL/kg/day
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
mL/kg/day | 1.36 [1.23 to 1.42]

6. Secondary Outcome: Study Part 1 (IV): Terminal Half-life
Description: Computed from the regression slope in the terminal phase of the model (the slope is biphasic). Terminal half life is the time it takes for the plasma concentration or the amount of immunoglobulin in the body to be reduced by 50%during the terminal phase.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
days | 33.1 [28.7 to 41.4]

7. Secondary Outcome: Study Part 2 (Subcutaneous (SC)): Maximum Plasma Concentration (C-max)
Description: Maximal immune globulin concentration after infusion
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: Participants for whom the following PK measurements are available: 1. pre-infusion and the Day 7 measurements 2. ≥2 measurements for Days 1, 3, and 5
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 31
g/L | 14.5 [12.3 to 16.4]

8. Secondary Outcome: Study Part 2 (SC): Time to Maximum Immune Globulin Concentration (T-max)
Description: Time to reach C-max
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 31
days | 4.8 [3.0 to 4.9]

9. Secondary Outcome: Study Part 2 (SC): Minimum Plasma Concentration (C-min)
Description: Minimal immune globulin concentration after infusion
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 31
g/L | 12.5 [11.3 to 14.2]

10. Secondary Outcome: Study Part 2 (SC): Weight-adjusted Clearance
Description: Computed as weight-adjusted dose divided by total AUC
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: mL/kg/day
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 31
mL/kg/day | 1.86 [1.61 to 2.04]

11. Secondary Outcome: Study Part 3B: Maximum Plasma Concentration (C-max)
Description: Maximal immune globulin concentration after infusion
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
g/L | 14.1 [12.5 to 16.3]

12. Secondary Outcome: Study Part 3B: Time to Maximum Immune Globulin Concentration (T-max)
Description: Time to reach C-max
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
days | 2.9 [1.2 to 3.2]

13. Secondary Outcome: Study Part 3B: Minimum Plasma Concentration (C-min)
Description: Minimal immune globulin concentration after infusion
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
g/L | 12.6 [10.6 to 14.0]

14. Secondary Outcome: Study Part 3B: Area Under the Curve (AUC)
Description: The AUC between adjacent infusions was calculated by the trapezoidal rule. Linear interpolation/extrapolation was used to calculate the AUC for the exact duration of the infusion intervals (21 or 28 days for IV administration and 7 days for SC administration). To allow for comparisons between Study Parts 1, 2 and 3b, AUC(0-τ) was standardized for the infusion intervals (3 or 4 weeks vs. 1 week).
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: g*days/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
g*days/L | 94.6 [80.4 to 106.9]

15. Secondary Outcome: Study Part 3B: Weight-adjusted Clearance
Description: Computed as weight-adjusted dose divided by total AUC
Time Frame: Pharmacokinetic evaluations: 60 minutes pre-infusion (before infusion #8 starts) up to 7 days (+/-1 day) post-infusion.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: mL/kg/day
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 32
mL/kg/day | 2.00 [1.84 to 2.12]

16. Secondary Outcome: Trough Levels of IgG After Administration of IGIV, 10%, in Participants 12 Years and Older
Description: Part 1: IgG trough levels measured at each IV infusion day (every 3rd or 4th week depending on schedule/frequency of participants for a total of 12 weeks) Part 2: IgG trough levels measured at weeks 1, 5 and 9 (of a total of 12 weeks) Part 3a: IgG trough levels measured at weeks 1 and 5 (of a total of 6 weeks) Part 3b: IgG trough levels measured at weeks 1, 5, 9 and 12 (of a total of 12 weeks)
Time Frame: as for outcome 2
Population: Full safety data set (all participants who received any study drug), 12 Years and Older
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | 12 Years and Older
Number analyzed (Participants) | 35
g/L
  Part 1, Screening visit (n=35) | 11.800 [10.300 to 13.000]
  Part 1, 3 week Interval, Visit 1 (n=4) | 10.900 [NA to NA] — Evaluable sample size was too small
  Part 1, 3 week Interval, Visit 2 (n=4) | 11.050 [NA to NA] — Evaluable sample size was too small
  Part 1, 3 week Interval, Visit 3 (n=5) | 14.000 [NA to NA] — Evaluable sample size was too small
  Part 1, 3 week Interval, Visit 4 (n=5) | 11.700 [NA to NA] — Evaluable sample size was too small
  Part 1, 3 week Interval, Visit 5 (n=5) | 12.400 [NA to NA] — Evaluable sample size was too small
  Part 1, 4 week Interval, Visit 1 (n=29) | 11.000 [10.000 to 12.300]
  Part 1, 4 week Interval, Visit 2 (n=29) | 10.800 [9.650 to 12.500]
  Part 1, 4 week Interval, Visit 3 (n=30) | 10.200 [9.480 to 12.600]
  Part 1, 4 week Interval, Visit 4 (n=30) | 10.150 [9.480 to 12.200]
  Part 2, Visit 1 (n=35) | 15.300 [14.800 to 17.100]
  Part 2, Visit 5 (n=34) | 12.700 [11.600 to 15.200]
  Part 2, Visit 9 (n=32) | 12.900 [11.800 to 14.800]
  Part 3a, Visit 1 (n=32) | 12.850 [11.600 to 14.900]
  Part 3a, Visit 5 (n=31) | 13.100 [11.400 to 15.100]
  Part 3b, Visit 1 (n=31) | 12.900 [11.600 to 15.200]
  Part 3b, Visit 5 (n=28) | 13.400 [11.000 to 14.600]
  Part 3b, Visit 9 (n=31) | 13.600 [11.000 to 14.400]
  End of Study (n=34) | 13.100 [11.300 to 14.400]

17. Secondary Outcome: Trough Levels of Antibody to Haemophilus Influenzae In All Study Participants
Description: Trough levels for IV and SC Treatment in Study Parts 1, 2, 3a and 3b.
Time Frame: Baseline; at each 3 or 4-week study visit in Study Part 1; at Visits 1, 5, and 9 in Study Part 2; at Visit 1 in Study Part 3a; at Visits 1, 5, and 9 in Study Part 3b; at Visit 1 in the Study Extension Part; and at the end-of-study evaluation
Population: All participants with specific antibody test results
Measure: Median (95% Confidence Interval); unit: µg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 49
µg/mL
  Part 1, Screening visit (n=49) | 2.790 [2.300 to 3.240]
  Part 1, 3 week Interval, Visit 1 (n=10) | 2.830 [2.020 to 4.350]
  Part 1, 3 week Interval, Visit 2 (n=10) | 2.885 [1.910 to 4.310]
  Part 1, 3 week Interval, Visit 3 (n=10) | 3.150 [2.030 to 3.950]
  Part 1, 3 week Interval, Visit 4 (n=10) | 3.145 [0.820 to 4.040]
  Part 1, 3 week Interval, Visit 5 (n=10) | 3.045 [1.650 to 4.140]
  Part 1, 4 week Interval, Visit 1 (n=38) | 2.210 [1.860 to 2.480]
  Part 1, 4 week Interval, Visit 2 (n=39) | 2.030 [1.680 to 2.780]
  Part 1, 4 week Interval, Visit 3 (n=39) | 2.130 [1.750 to 2.670]
  Part 1, 4 week Interval, Visit 4 (n=38) | 2.135 [2.020 to 2.610]
  Part 2, Visit 1 (n=47) | 3.280 [3.000 to 3.860]
  Part 2, Visit 5 (n=46) | 2.810 [2.360 to 3.080]
  Part 2, Visit 9 (n=44) | 3.175 [2.530 to 3.470]
  Part 3a, Visit 1 (n=44) | 2.840 [2.400 to 3.160]
  Part 3b, Visit 1 (n=43) | 3.030 [2.610 to 3.500]
  Part 3b, Visit 5 (n=41) | 3.070 [2.820 to 3.650]
  Part 3b, Visit 9 (n=44) | 3.285 [2.780 to 3.870]
  Extension, Visit 1 (n=36) | 2.940 [2.530 to 3.780]
  End of Study (n=46) | 3.010 [2.660 to 3.690]

18. Secondary Outcome: Trough Levels of Antibody to Hepatitis B in All Study Participants
Description: Trough levels for IV and SC Treatment in Study Parts 1, 2, 3a and 3b.
Time Frame: as for outcome 17
Population: All participants with specific antibody test results
Measure: Median (95% Confidence Interval); unit: mIU/mL
Arm/Group | All Participants
Number analyzed (Participants) | 49
mIU/mL
  Part 1, Screening visit (n=36) | 239.450 [180.000 to 293.300]
  Part 1, 3 week Interval, Visit 1 (n=8) | 182.050 [139.500 to 789.000]
  Part 1, 3 week Interval, Visit 2 (n=10) | 251.150 [208.600 to 311.900]
  Part 1, 3 week Interval, Visit 3 (n=10) | 282.050 [231.900 to 333.900]
  Part 1, 3 week Interval, Visit 4 (n=10) | 274.200 [223.100 to 460.700]
  Part 1, 3 week Interval, Visit 5 (n=10) | 261.850 [233.900 to 292.400]
  Part 1, 4 week Interval, Visit 1 (n=36) | 197.750 [135.600 to 242.200]
  Part 1, 4 week Interval, Visit 2 (n=39) | 213.600 [191.000 to 282.500]
  Part 1, 4 week Interval, Visit 3 (n=39) | 202.800 [172.200 to 262.600]
  Part 1, 4 week Interval, Visit 4 (n=38) | 207.850 [183.800 to 265.800]
  Part 2, Visit 1 (n=46) | 401.350 [380.800 to 482.200]
  Part 2, Visit 5 (n=46) | 341.100 [301.700 to 364.700]
  Part 2, Visit 9 (n=44) | 316.800 [282.800 to 367.900]
  Part 3a, Visit 1 (n=44) | 318.450 [280.200 to 351.000]
  Part 3b, Visit 1 (n=43) | 385.200 [304.300 to 454.300]
  Part 3b, Visit 5 (n=41) | 314.100 [247.200 to 374.900]
  Part 3b, Visit 9 (n=44) | 351.050 [292.000 to 412.200]
  Extension, Visit 1 (n=36) | 328.750 [273.100 to 368.400]
  End of Study (n=44) | 319.600 [297.000 to 372.400]

19. Primary Outcome: Percentage of Participants in Full Safety Data Set (FSDS) Who Had Any Infusion for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped
Description: Ability to tolerate IGIV, 10% administered IV or SC. Measured as the percentage of participants for which the infusion rate was reduced at any infusion and/or the infusion was interrupted or stopped for (i) any reason and (ii) for tolerability concerns or AEs
Time Frame: Throughout study (1 year and 9 months)
Population: Full safety data set (all participants who received any study drug)
Measure: Number; unit: Percentage of Participants
Groups:
- Infusion Rate Change - For Any Reason: Infusion Rate Reduced and/or Infusion Interrupted or Stopped for Any Reason
- Infusion Rate Change - For Tolerability/AE: Infusion Rate Reduced and/or Infusion Interrupted or Stopped for Tolerability/AEs
Arm/Group | Infusion Rate Change - For Any Reason | Infusion Rate Change - For Tolerability/AE
Number analyzed (Participants) | 49 | 49
Percentage of Participants
  Study Part 1 (IV) (n= 49) | 18.4 | 16.3
  Study Part 2 (SC) (n= 47) | 29.8 | 4.3
  Study Part 3A (SC) (n=44) | 15.9 | 2.3
  Study Part 3B (SC) (n=44) | 13.6 | 2.3
  Study Extension (SC) (n= 36) | 13.9 | 0.0
  Study Part 2, 3A, 3B, Study Extension (n= 47) | 40.4 | 4.3

20. Secondary Outcome: Trough Levels of Antibody to Tetanus In All Study Participants
Description: Trough levels for IV and SC Treatment in Study Parts 1, 2, 3a and 3b.
Time Frame: as for outcome 17
Population: All participants with specific antibody test results
Measure: Median (95% Confidence Interval); unit: IU/mL
Arm/Group | All Participants
Number analyzed (Participants) | 49
IU/mL
  Part 1, Screening visit (n=49) | 2.840 [2.500 to 3.660]
  Part 1, 3 week Interval, Visit 1 (n=10) | 3.010 [1.740 to 3.640]
  Part 1, 3 week Interval, Visit 2 (n=10) | 3.500 [1.970 to 4.640]
  Part 1, 3 week Interval, Visit 3 (n=10) | 3.360 [2.180 to 4.540]
  Part 1, 3 week Interval, Visit 4 (n=10) | 3.205 [1.810 to 5.030]
  Part 1, 3 week Interval, Visit 5 (n=10) | 3.520 [2.230 to 4.220]
  Part 1, 4 week Interval, Visit 1 (n=37) | 2.340 [1.980 to 2.830]
  Part 1, 4 week Interval, Visit 2 (n=39) | 2.360 [1.880 to 2.760]
  Part 1, 4 week Interval, Visit 3 (n=38) | 2.125 [1.890 to 2.680]
  Part 1, 4 week Interval, Visit 4 (n=36) | 2.325 [1.910 to 2.800]
  Part 2, Visit 1 (n=47) | 4.310 [3.890 to 5.050]
  Part 2, Visit 5 (n=46) | 3.445 [2.920 to 4.030]
  Part 2, Visit 9 (n=43) | 3.720 [3.090 to 4.160]
  Part 3a, Visit 1 (n=44) | 3.090 [2.670 to 3.830]
  Part 3b, Visit 1 (n=43) | 3.690 [3.210 to 4.220]
  Part 3b, Visit 5 (n=41) | 3.410 [2.780 to 4.440]
  Part 3b, Visit 9 (n=43) | 3.150 [2.920 to 3.920]
  Extension, Visit 1 (n=36) | 3.355 [2.440 to 4.480]
  End of Study (n=46) | 3.860 [3.150 to 5.000]

21. Secondary Outcome: Number of Anti-Measles Antibody Titers That Were Below or Above the Protective Titer Level
Description: Antibody Titers That Were Below or Above the Protective Titer Level of >1:8 for IV and SC Treatment in Study Parts 1, 2, 3a and 3b. Participants had multiple anti-measles antibody titers measured during the study.
Time Frame: as for outcome 17
Population: All study participants
Measure: Number; unit: Antibody titers
Units Other Than Participants: Antibody titers
Arm/Group | Full Safety Data Set
Number analyzed (Participants) | 49
Number analyzed (Antibody titers) | 654
Antibody titers
  Anti-Measles Antibody Tests Below a Titer of >1:8 | 0
  Anti-Measles Antibody Tests Above a Titer of >1:8 | 654

22. Secondary Outcome: Annual Infection Rates During Treatment
Description: Annual rate of all infections calculated using a Poisson model to account for different lengths of observation per subject using SAS V9.1.3 procedure GENMOD with allowance for overdispersion by deviance method. Point estimates and likelihood-ratio based 95% confidence intervals were provided. Infections as included in analysis comprised all reported AEs that were coded to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) of infections and infestations, described as an infection by investigator, or for which anti-infective medication was prescribed.
Time Frame: Throughout the study, 1 year and 9 months
Population: Full safety data set (all participants who received any study drug)
Measure: Mean (95% Confidence Interval); unit: Estimated infections per year
Arm/Group | 2 to <12 Years | 12 Years and Older
Number analyzed (Participants) | 14 | 35
Estimated infections per year
  Study Part 1 (IV) | 5.0 [2.3 to 9.3] | 5.2 [3.6 to 7.2]
  Study Part 2 (SC) | 5.6 [2.7 to 10.0] | 4.1 [2.6 to 6.1]
  Study Part 3A (SC) | 3.5 [1.4 to 7.1] | 4.6 [2.6 to 7.3]
  Study Part 3B (SC) | 3.9 [1.6 to 7.8] | 3.8 [2.4 to 5.8]
  Study Extension (SC) | 4.0 [2.4 to 6.2] | 3.8 [2.6 to 5.3]
  Study Part 2, 3A, 3B, Study Extension (all SC) | 4.3 [2.8 to 6.4] | 4.0 [3.0 to 5.2]

23. Secondary Outcome: Annual Rate of Acute Serious Bacterial Infections During IV and SC Treatment (FSDS)
Description: Annual rate of validated acute serious bacterial infections was calculated using a Poisson model to account for the different lengths of observation per subject using SAS V9.1.3 procedure GENMOD with an allowance for overdispersion by the deviance method.
Time Frame: Throughout the study, 1 year and 9 months
Population: Full Safety Data Set (All study participants who received any infusions)
Measure: Number; unit: Estimated infections/year
Groups:
- IV Treatment: Study Part 1
- All SC Treatment Periods: Study Parts 2, 3a, 3b, extension
Arm/Group | IV Treatment | All SC Treatment Periods
Number analyzed (Participants) | 49 | 47
Estimated infections/year | 0.000 | 0.067
Statistical Analysis 1: Comparison: All SC Treatment Periods; Test type: Superiority or Other; Poisson = 0.067, 99% CI 1-sided [upper limit 0.134]

24. Secondary Outcome: Rate of Temporally Associated AEs Per Infusion
Description: Rate of AEs per infusion defined as the total number of all AEs that begin during infusion or within 72 hours of completion of an infusion ("temporally associated") divided by the total number of infusions.
Time Frame: During Infusion or Within 72 Hours of Completion of Infusions
Population: All participants who received any study drug
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Groups:
- FSDS: All participants who received any study drug
- SNSC: Dataset of subjects naïve to SC administration of immunoglobulins
- SESC: Dataset of subjects with prior experience with subcutaneous administration of immunoglobulins
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
AEs per infusion
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 0.25 | 0.45 | 0.00
  Study Part 2 (SC) (N = 595, 469, 126) | 0.08 | 0.13 | 0.08
  Study Part 3a (SC) (N = 268, 206, 62) | 0.00 | 0.08 | 0.00
  Study Part 3b (SC) (N = 538, 418, 120) | 0.08 | 0.08 | 0.00
  Study Extension (SC) (N = 893, 664, 229) | 0.07 | 0.09 | 0.00
  Total SC (N = 2294, 1757, 537) | 0.08 | 0.08 | 0.00

25. Secondary Outcome: AEs Deemed/Judged to be Related by the Investigator
Description: Rate of related AEs defined as the total number of AEs determined by the investigator to be related to the study drug that occur at any time during the study divided by the total number of infusions.
Time Frame: Throughout the study period (1 year and 9 months)
Population: All participants who received any study drug
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Groups:
- SNSC: Dataset of participants naïve to SC administration of immunoglobulins
- SESC: Dataset of participants with prior experience with subcutaneous administration of immunoglobulins
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
AEs per infusion
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 0.00 | 0.25 | 0.00
  Study Part 2 (SC) (N = 595, 469, 126) | 0.07 | 0.06 | 0.08
  Study Part 3a (SC) (N = 268, 206, 62) | 0.00 | 0.00 | 0.00
  Study Part 3b (SC) (N = 538, 418, 120) | 0.00 | 0.00 | 0.00
  Study Extension (SC) (N = 893, 664, 229) | 0.00 | 0.03 | 0.00
  Total SC (Study Parts 2, 3A, 3B, Study Extension) | 0.00 | 0.00 | 0.00

26. Secondary Outcome: Frequency of Dose Adjustments (If IgG Trough Levels <4.5 g/L)
Description: Frequency of Dose Adjustments Based on IgG Trough Levels <4.5 g/L IgG, if Any, for Each Study Part. Defined/calculated as the number of participants requiring dose adjustments divided by the number of participants, for each respective data set.
Time Frame: Throughout the study period (1 year and 9 months)
Population: All participants who received any study drug
Measure: Number; unit: ratio
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
ratio
  Study Part 1 (IV) | 0.00 | 0.00 | 0.00
  Study Part 2 (SC) | 0.00 | 0.00 | 0.00
  Study Part 3a (SC) | 0.00 | 0.00 | 0.00
  Study Part 3b (SC) | 0.00 | 0.00 | 0.00
  Study Extension (SC) | 0.00 | 0.00 | 0.00
  Total SC (Study Parts 2, 3A, 3B, Study Extension) | 0.00 | 0.00 | 0.00

27. Secondary Outcome: Proportion of Participants Reporting ≥1 Temporally Associated Moderate or Severe AEs
Description: Proportion of Participants Reporting 1 or More Moderate or Severe AEs That Begin During Infusion or Within 72 Hours of Completion of an Infusion.
Time Frame: During Infusion or Within 72 Hours of Completion of Infusions
Population: All participants who received any study drug
Measure: Number; unit: Proportion of participants
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Proportion of participants
  Study Part 1 (IV) | 0.43 | 0.47 | 0.27
  Study Part 2 (SC) | 0.36 | 0.44 | 0.09
  Study Part 3a (SC) | 0.23 | 0.24 | 0.20
  Study Part 3b (SC) | 0.36 | 0.38 | 0.30
  Study Extension (SC) | 0.50 | 0.56 | 0.33
  Total SC (Study Parts 2, 3A, 3B, Study Extension) | 0.66 | 0.75 | 0.36

28. Primary Outcome: Percentage of Participants Naïve to SC Administration of Immunoglobulins (SNSC) Who Had Any Infusion for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped.
Description: as for outcome 19
Time Frame: Throughout study (1 year and 9 months)
Population: SNSC data set (all participants naïve to SC administration of immunoglobulins who received any study drug)
Measure: Number; unit: Percentage of Participants
Arm/Group | Infusion Rate Change - For Any Reason | Infusion Rate Change - For Tolerability/AE
Number analyzed (Participants) | 38 | 38
Percentage of Participants
  Study Part 1 (IV) (n= 38) | 23.7 | 21.1
  Study Part 2 (SC) (n= 36) | 33.3 | 5.6
  Study Part 3A (SC) (n=34) | 20.6 | 2.9
  Study Part 3B (SC) (n=34) | 17.6 | 2.9
  Study Extension (SC) (n= 27) | 14.8 | 0.0
  Study Part 2, 3A, 3B, Study Extension (n= 36) | 47.2 | 5.6

29. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Severity, and Causality (FSDS)
Description: Seriousness and causality are abbreviated below as: Seriousness: Serious Adverse Event= SAE, non-Serious Adverse Event= non-SAE Causality: possibly or probably related= R, not related= NR
Time Frame: Throughout entire study (1 year and 9 months)
Population: All study participants who received any study drug during each of the study parts
Measure: Number; unit: Adverse events
Arm/Group | Study Part 1, IV Administration | Study Part 2, SC Administration | Study Part 3a, SC Administration | Study Part 3b, SC Administration | Study Extension, SC Administration | Total SC (Parts 2, 3a, 3b, Extension)
Number analyzed (Participants) | 49 | 47 | 44 | 44 | 36 | 47
Adverse events
  Abdominal Discomfort- non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 3 | 3
  Abdominal Distension-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 7 | 7
  Abdominal Distension-non-SAE, NR, Moderate | 0 | 0 | 0 | 2 | 2 | 4
  Abdominal Distension-non-SAE, R, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Abdominal Distension-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Abdominal Pain-non-SAE, NR, Mild | 1 | 0 | 1 | 0 | 1 | 2
  Abdominal Pain-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Abdominal Pain Upper-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 6 | 6
  Abdominal Pain Upper-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Abdominal Pain Upper-non-SAE, R, Mild | 0 | 3 | 1 | 0 | 0 | 4
  Abdominal Tenderness-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Acne-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Acne-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Acute Sinusitis-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Addison's Disease-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Addison's Disease-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Alopecia-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Ammonia Increased-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Animal Bite-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Anorexia-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Anxiety-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Aphthous Stomatitis-non-SAE, NR, Mild | 0 | 1 | 1 | 0 | 2 | 4
  Arthralgia-non-SAE, NR, Moderate | 0 | 3 | 1 | 2 | 1 | 7
  Arthralgia-non-SAE, NR, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Arthralgia-non-SAE, R, Mild | 1 | 0 | 1 | 0 | 0 | 1
  Arthralgia-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Arthritis-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Arthropod Bite-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 1 | 2
  Asthenia-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Asthenia-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Asthma-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Asthma-non-SAE, NR, Moderate | 3 | 0 | 1 | 1 | 3 | 5
  Asthma-non-SAE, NR, Severe | 0 | 0 | 0 | 1 | 0 | 1
  Asthma-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Asthma Exercise Induced-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  ADHD-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Back Pain-non-SAE, NR, Mild | 1 | 0 | 0 | 2 | 0 | 2
  Back Pain-non-SAE, NR, Moderate | 1 | 0 | 0 | 2 | 0 | 2
  Back Pain-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Biliary Tract Infection Bacterial-SAE, NR, Moderat | 0 | 1 | 0 | 0 | 0 | 1
  Blepharitis-non-SAE,NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Blepharitis-non-SAE,NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  B.P. Diastolic Decreased-non-SAE, R, Mild | 0 | 0 | 2 | 0 | 0 | 2
  Blood Pressure Increased-non-SAE, NR, Mild | 0 | 0 | 0 | 2 | 0 | 2
  Blood Pressure Increased-non-SAE, R, Mild | 0 | 0 | 0 | 1 | 0 | 1
  B.P. Systolic Increased-non-SAE, NR, Mild | 0 | 1 | 1 | 0 | 0 | 2
  B.P. Systolic Increased-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  B.P. Systolic Increased-non-SAE, R, Mild | 1 | 4 | 2 | 0 | 0 | 6
  B.P. Systolic Increased-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Breast Tenderness-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Breath Sounds Abnormal-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Bronchitis-non-SAE, NR, Mild | 1 | 1 | 0 | 2 | 2 | 5
  Bronchitis-non-SAE, NR, Moderate | 1 | 0 | 1 | 0 | 4 | 5
  Bursitis-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Candidiasis-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Cardiac Murmur-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Centrl Venous Catheterisation-non-SAE, NR, Moderat | 0 | 0 | 0 | 0 | 1 | 1
  Cervical Spinal Stenosis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Chest Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Chest Pain-SAE, NR, Severe | 0 | 0 | 0 | 1 | 0 | 1
  Chills-non-SAE, R, Mild | 7 | 0 | 0 | 0 | 0 | 0
  Chills-non-SAE, R, Moderate | 6 | 0 | 0 | 0 | 0 | 0
  C.O.P.D.-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  C.O.P.D.-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Chronic Sinusitis-non-SAE, NR, Mild | 0 | 0 | 1 | 2 | 1 | 4
  Chronic Sinusitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Confusional State-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Conjunctival Hyperaemia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Conjunctivitis Allergic-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Conjunctivitis Bacterial-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Conjunctivitis Infective-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Conjunctivitis Infective-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Constipation-non-SAE, NR, Mild | 1 | 2 | 0 | 0 | 1 | 3
  Constipation-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Contusion-non-SAE, NR, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Contusion-non-SAE, R, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Convulsion-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Convulsion-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Costochondritis-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Costochondritis-non-SAE, NR, Severe | 0 | 1 | 0 | 0 | 0 | 1
  Cough-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 2 | 2
  Cough-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Croup Infectious-non-SAE, NR, Mild | 0 | 2 | 0 | 1 | 0 | 3
  Croup Infectious-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Cryptosporidiosis Infection-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Cystitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Dental Caries-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Dermatitis-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Dermatitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dermatitis Contact-non-SAE, NR, Moderate | 1 | 1 | 1 | 1 | 0 | 3
  Device Failure-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Diarrhoea-non-SAE, NR, Mild | 1 | 2 | 0 | 2 | 2 | 6
  Diarrhoea-non-SAE, NR, Moderate | 2 | 2 | 1 | 1 | 0 | 4
  Diarrhoea-non-SAE, R, Mild | 0 | 0 | 2 | 0 | 1 | 3
  Diarrhoea Haemorrhagic-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Diarrhoea Infectious-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Diverticulitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Drug Eruption-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dyspepsia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Dyspnoea-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Dyspnoea-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Dyspnoea-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Ear Infection-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 1 | 1
  Ear Pain-non-SAE, NR, Mild | 1 | 1 | 1 | 0 | 2 | 4
  Ear Pain-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Eczema-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 3 | 4
  Eczema-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Epistaxis-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Epistaxis-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 1 | 2
  Excoriation-non-SAE, NR, Mild | 0 | 0 | 0 | 2 | 0 | 2
  Exostosis-non-SAE, NR,Mild | 0 | 0 | 1 | 0 | 0 | 1
  Eye Infection Viral-non-SAE, NR, Moderate | 3 | 1 | 0 | 2 | 1 | 4
  Eye Irritation-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Eye Oedema-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Fall-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Fatigue-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Fatigue-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Fatigue-non-SAE, R, Mild | 1 | 4 | 0 | 2 | 0 | 6
  Fatigue-non-SAE, R, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Flank Pain-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Flatulence-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Flatulence-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Folliculitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Fungal Infection-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Furuncle-non-SAE, NR, Moderate | 0 | 1 | 1 | 0 | 0 | 2
  Gastric Ulcer-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Gastric Ulcer-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Gastroenteritis-non-SAE, NR, Mild | 1 | 0 | 0 | 1 | 0 | 1
  Gastroenteritis-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Gastroenteritis-non-SAE, R, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Gastroenteritis Viral-non-SAE, NR, Mild | 2 | 2 | 0 | 0 | 0 | 2
  Gastroenteritis Viral-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 3 | 4
  Goitre-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Gravitational Oedema-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Haematochezia-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Haemoglobin Decreased-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Haemorrhoids-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Head Injury-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Headache-non-SAE, NR, Mild | 8 | 5 | 3 | 4 | 8 | 20
  Headache-non-SAE, NR, Moderate | 4 | 0 | 2 | 1 | 1 | 4
  Headache-non-SAE, NR, Severe | 0 | 0 | 1 | 0 | 1 | 2
  Headache-non-SAE, R, Mild | 19 | 6 | 1 | 2 | 8 | 17
  Headache-non-SAE, R, Moderate | 8 | 1 | 1 | 0 | 0 | 2
  Headache-non-SAE, R, Severe | 3 | 1 | 0 | 0 | 0 | 1
  Heart Rate Decreased-non-SAE, R, Mild | 0 | 0 | 3 | 0 | 0 | 3
  Heart Rate Increased-non-SAE, NR, Mild | 0 | 3 | 0 | 1 | 0 | 4
  Heart Rate Increased-non-SAE, R, Mild | 4 | 4 | 3 | 1 | 1 | 9
  Heart Rate Increased-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Hiatus Hernia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Hordeolum-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Hyperlipidaemia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Hypoxia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Implant Site Pain-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Infection-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 1 | 1
  Infection-non-SAE, NR, Moderate | 1 | 1 | 1 | 0 | 1 | 3
  Influenza-non-SAE, NR, Mild | 1 | 3 | 0 | 0 | 2 | 5
  Influenza-non-SAE, NR, Moderate | 2 | 4 | 0 | 1 | 2 | 7
  Infusion Related Reaction-non-SAE, R, Mild | 1 | 1 | 0 | 0 | 0 | 1
  Infusion Site Erythema-non-SAE, R, Mild | 0 | 3 | 0 | 0 | 0 | 3
  Infusion Site Haematoma-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 1 | 2
  Infusion Site Haematoma-non-SAE, R, Mild | 0 | 2 | 2 | 2 | 6 | 12
  Infusion Site Haematoma-non-SAE, R, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Infusion Site Haemorrhage-non-SAE, R, Mild | 0 | 2 | 0 | 0 | 0 | 2
  Infusion Site Irritation-non-SAE, R, Mild | 1 | 1 | 0 | 0 | 1 | 2
  Infusion Site Oedema-non-SAE, R, Mild | 0 | 3 | 0 | 0 | 0 | 3
  Infusion Site Pain-non-SAE, R, Mild | 1 | 9 | 2 | 2 | 1 | 14
  Infusion Site Pain-non-SAE, R, Moderate | 0 | 5 | 1 | 2 | 0 | 8
  Infusion Site Pruritus-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Pruritus-non-SAE, R, Mild | 0 | 2 | 1 | 1 | 0 | 4
  Infusion Site Pruritus-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Rash-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Rash-non-SAE, R, Mild | 0 | 1 | 1 | 0 | 1 | 3
  Infusion Site Reaction-non-SAE, R, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Infusion Site Swelling-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Swelling-non-SAE, R, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Infusion Site Vesicles-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Inguinal Mass-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Injection Site Haematoma-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Injection Site Haematoma-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Injection Site Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Insomnia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 2 | 3
  Insomnia-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Intermit. Explosive Disorder-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Irritability-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Irritable Bowel Syndrome-non-SAE, NR, Moderate | 0 | 1 | 0 | 1 | 1 | 3
  Joint Dislocation-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Joint Sprain-non-SAE, NR, Mild | 0 | 2 | 0 | 0 | 0 | 2
  Joint Swelling-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Joint Swelling-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Laryngitis-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Laryngitis-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Laryngitis Viral-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Lethargy-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Limb Injury-non-SAE, NR, Mild | 1 | 0 | 0 | 1 | 0 | 1
  Lip Ulceration-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Livedo Reticularis-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Lung Infection-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Lung Infection-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Lymphadenopathy-non-SAE, NR, Mild | 2 | 0 | 1 | 0 | 2 | 3
  Malaise-non-SAE, NR, Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Malaise-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Memory Impairment-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Middle Ear Effusion-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Migraine-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 1 | 2
  Migraine-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Migraine-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Migraine-non-SAE, R, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Migraine-non-SAE, R, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Mouth Ulceration-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Muscle Strain-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 1 | 2
  Muscular Weakness-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Musculoskeletal Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Musculoskeletal Pain-non-SAE, NR, Moderate | 0 | 0 | 1 | 1 | 1 | 3
  Myalgia-non-SAE, NR, Mild | 0 | 1 | 1 | 1 | 5 | 8
  Myalgia-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Myopia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Nasal Congestion-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Nasal Congestion-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 1 | 2
  Nasal Disorder-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Nasal Mucosal Disorder-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Nasal Polyps-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Nasopharyngitis-non-SAE, NR, Mild | 5 | 1 | 0 | 1 | 4 | 6
  Nasopharyngitis-non-SAE, NR, Moderate | 0 | 1 | 0 | 1 | 4 | 6
  Nausea-non-SAE, NR, Mild | 1 | 3 | 1 | 2 | 5 | 11
  Nausea-non-SAE, NR, Moderate | 0 | 1 | 0 | 2 | 1 | 4
  Nausea-non-SAE, NR, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Nausea-non-SAE, R, Mild | 4 | 1 | 1 | 3 | 1 | 6
  Nausea-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Oedema Peripheral-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Oedema Peripheral-non-SAE, R, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Oral Herpes-non-SAE, NR, Mild | 0 | 3 | 0 | 0 | 1 | 4
  Oropharyngeal Pain-non-SAE, NR, Mild | 1 | 2 | 0 | 0 | 3 | 5
  Oropharyngeal Pain-non-SAE, NR, Moderate | 2 | 0 | 0 | 1 | 2 | 3
  Osteomyelitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Osteopenia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Otitis Externa-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Otitis Media-non-SAE, NR, Mild | 0 | 3 | 1 | 0 | 0 | 4
  Otitis Media-non-SAE, NR, Moderate | 0 | 2 | 0 | 3 | 2 | 7
  Pain-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Pain In Extremity-non-SAE, NR, Mild | 3 | 0 | 0 | 0 | 0 | 0
  Pain In Extremity-non-SAE, NR, Moderate | 0 | 0 | 1 | 1 | 0 | 2
  Pain In Extremity-non-SAE, R, Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Pain In Extremity-non-SAE, R, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Paraesthesia-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Paronychia-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Periorbital Oedema-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Pharyngitis-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 1 | 2
  Pharyngitis-non-SAE, NR, Moderate | 2 | 1 | 0 | 2 | 0 | 3
  Pharyngitis Streptococcal-non-SAE, NR, Moderate | 0 | 2 | 0 | 0 | 0 | 2
  Pneumonia-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Pneumonia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 2 | 3
  Pneumonia Bacterial-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Pneumonia Streptococcal-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Procedural Pain-non-SAE, NR, Moderate | 1 | 0 | 0 | 1 | 2 | 3
  Pyrexia-non-SAE, NR, Mild | 1 | 3 | 0 | 0 | 10 | 13
  Pyrexia-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 2 | 2
  Pyrexia-non-SAE, R, Mild | 5 | 2 | 0 | 0 | 4 | 6
  Pyrexia-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 1 | 1
  Rales-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Rash-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Rash-non-SAE, R, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Rash Erythematous-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 1 | 2
  Rash Macular-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Rash Papular-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Rash Pruritic-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Respiratory Rate Increased-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Respir. Tract Infect. Viral-non-SAE, NR, Mild | 2 | 2 | 0 | 0 | 1 | 3
  Respir. Tract Infect Viral-non-SAE, NR, Moderate | 1 | 1 | 0 | 0 | 0 | 1
  Rhinitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Rhinitis Allergic-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Rhinorrhoea-non-SAE, NR, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Road Traffic Accident-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Scleritis-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Scleritis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Scoliosis-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Sinus Congestion-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 1 | 1
  Sinus Congestion-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Sinus Disorder-non-SAE, NR, Severe | 0 | 1 | 0 | 0 | 0 | 1
  Sinus Headache-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 1 | 1
  Sinus Headache-non-SAE, NR, Moderate | 2 | 1 | 0 | 1 | 0 | 2
  Sinusitis-non-SAE, NR, Mild | 3 | 0 | 0 | 1 | 4 | 5
  Sinusitis-non-SAE, NR, Moderate | 7 | 4 | 6 | 5 | 3 | 18
  Sinusitis-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Sinusitis Fungal-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Skin Laceration-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Skin Lesion-non-SAE, NR, Mild | 1 | 0 | 0 | 1 | 0 | 1
  Skin Papilloma-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Skin Warm-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Sports Injury-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Streptococcal Infection-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Subcutaneous Abscess-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Suicidal Ideation-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Sunburn-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Tendonitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Tooth Fracture-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Tooth Infection-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Toothache-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 1 | 2
  Tourette's Disorder-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Upper Respir. Tract Congestion-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Upper Respir. Tract Infection-non-SAE, NR, Mild | 4 | 3 | 3 | 6 | 8 | 20
  Upper Respir. Tract Infect.-non-SAE, NR, Moderate | 2 | 1 | 0 | 1 | 3 | 5
  Urinary Tract Infection-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 1 | 1
  Urticaria-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Urticaria-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Vaginal Lesion-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Vaginitis Bacterial-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Varicose Vein-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Varicose Vein-non-SAE, NR, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Vestibulitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Viral Infection-non-SAE, NR, Mild | 2 | 2 | 0 | 0 | 0 | 2
  Viral Infection-non-SAE, NR, Moderate | 3 | 0 | 0 | 1 | 0 | 1
  Viral Skin Infection-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Viral Upper Respir. Tract Infect-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Viral Up. Respir Tract Infec-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Vitamin D Deficiency-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Vomiting-non-SAE, NR, Mild | 2 | 1 | 1 | 1 | 4 | 7
  Vomiting-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Vomiting-non-SAE, R, Mild | 8 | 0 | 0 | 1 | 1 | 2
  Vomiting-non-SAE, R, Moderate | 1 | 0 | 0 | 2 | 0 | 2
  Vulvovaginal Candidiasis-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Vulvovaginal Mycotic Infection-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Vulvovaginal Mycotic Infect.-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Wheezing-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Wound-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1

30. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Severity, and Causality (FSDS)
Description: Seriousness and causality are abbreviated below as: Seriousness: Serious Adverse Event= SAE, non-Serious Adverse Event= non-SAE Causality: possibly or probably related= R, not related= NR Rate of AEs defined as the number of AEs categorized by MedDRA preferred terms, seriousness, severity, and causality divided by the number of infusions.
Time Frame: Throughout entire study (1 year and 9 months)
Population: All study participants who received any study drug during each of the study parts
Measure: Number; unit: AEs per infusion
Arm/Group | Study Part 1, IV Administration | Study Part 2, SC Administration | Study Part 3a, SC Administration | Study Part 3b, SC Administration | Study Extension, SC Administration | Total SC (Parts 2, 3a, 3b, Extension)
Number analyzed (Participants) | 49 | 47 | 44 | 44 | 36 | 47
AEs per infusion
  Abdominal Discomfort- non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Abdominal Distension-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.29 | 0.29
  Abdominal Distension-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.17 | 0.08 | 0.13
  Abdominal Distension-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Abdominal Distension-non-SAE, R, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Abdominal Pain-non-SAE, NR, Mild | 0.25 | 0.00 | 0.17 | 0.00 | 0.05 | 0.11
  Abdominal Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Abdominal Pain Upper-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Abdominal Pain Upper-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.08 | 0.08
  Abdominal Pain Upper-non-SAE, R, Mild | 0.00 | 0.10 | 0.17 | 0.00 | 0.00 | 0.13
  Abdominal Tenderness-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Acne-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Acne-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Acute Sinusitis-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Addison's Disease-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Addison's Disease-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Alopecia-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Ammonia Increased-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Animal Bite-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Anorexia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Anxiety-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Aphthous Stomatitis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.14 | 0.14
  Arthralgia-non-SAE, NR, Moderate | 0.00 | 0.10 | 0.17 | 0.17 | 0.04 | 0.11
  Arthralgia-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Arthralgia-non-SAE, R, Mild | 0.25 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Arthralgia-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Arthritis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Arthropod Bite-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.03 | 0.06
  Asthenia-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Asthenia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Asthma-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Asthma-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.08 | 0.03 | 0.04
  Asthma-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Asthma-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Asthma Exercise Induced-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  ADHD-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Back Pain-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Back Pain-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.17 | 0.00 | 0.17
  Back Pain-non-SAE, R, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Biliary Tract Infection Bacterial-SAE, NR, Moderat | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Blepharitis-non-SAE,NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Blepharitis-non-SAE,NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  B.P. Diastolic Decreased-non-SAE, R, Mild | 0.00 | 0.00 | 0.33 | 0.00 | 0.00 | 0.33
  Blood Pressure Increased-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.17 | 0.00 | 0.17
  Blood Pressure Increased-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  B.P. Systolic Increased-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.00 | 0.12
  B.P. Systolic Increased-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  B.P. Systolic Increased-non-SAE, R, Mild | 0.25 | 0.16 | 0.17 | 0.00 | 0.00 | 0.17
  B.P. Systolic Increased-non-SAE, R, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Breast Tenderness-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Breath Sounds Abnormal-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Bronchitis-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.17 | 0.06 | 0.08
  Bronchitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.00 | 0.07 | 0.08
  Bursitis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Candidiasis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Cardiac Murmur-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Centrl Venous Catheterisation-non-SAE, NR, Moderat | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Cervical Spinal Stenosis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Chest Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Chest Pain-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Chills-non-SAE, R, Mild | 0.75 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Chills-non-SAE, R, Moderate | 0.75 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  C.O.P.D.-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  C.O.P.D.-non-SAE, NR, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Chronic Sinusitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.08 | 0.03 | 0.08
  Chronic Sinusitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Confusional State-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Conjunctival Hyperaemia-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Conjunctivitis Allergic-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Conjunctivitis Bacterial-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Conjunctivitis Infective-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Conjunctivitis Infective-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Constipation-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.03 | 0.07
  Constipation-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Contusion-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Contusion-non-SAE, R, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Convulsion-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Convulsion-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Costochondritis-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Costochondritis-non-SAE, NR, Severe | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Cough-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Cough-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Croup Infectious-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Croup Infectious-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.11 | 0.11
  Cryptosporidiosis Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Cystitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Dental Caries-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Dermatitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Dermatitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Dermatitis Contact-non-SAE, NR, Moderate | 0.25 | 0.08 | 0.17 | 0.08 | 0.00 | 0.08
  Device Failure-non-SAE, NR, Mild | 0.23 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Diarrhoea-non-SAE, NR, Mild | 0.25 | 0.07 | 0.00 | 0.17 | 0.05 | 0.06
  Diarrhoea-non-SAE, NR, Moderate | 0.25 | 0.17 | 0.17 | 0.08 | 0.00 | 0.17
  Diarrhoea-non-SAE, R, Mild | 0.00 | 0.00 | 0.33 | 0.00 | 0.05 | 0.19
  Diarrhoea Haemorrhagic-non-SAE, NR,Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Diarrhoea Infectious-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Diverticulitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Drug Eruption-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Dyspepsia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Dyspnoea-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Dyspnoea-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Dyspnoea-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Ear Infection-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Ear Pain-non-SAE, NR, Mild | 0.25 | 0.06 | 0.17 | 0.00 | 0.04 | 0.05
  Ear Pain-non-SAE, R, Moderate | 0.00 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Eczema-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.04 | 0.06
  Eczema-non-SAE, NR, Severe | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Epistaxis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Epistaxis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.14 | 0.00 | 0.07 | 0.10
  Excoriation-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.17 | 0.00 | 0.17
  Exostosis-non-SAE, NR,Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Eye Infection Viral-non-SAE, NR, Moderate | 0.38 | 0.10 | 0.00 | 0.08 | 0.04 | 0.08
  Eye Irritation-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Eye Oedema-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Fall-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Fatigue-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.11 | 0.11
  Fatigue-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Fatigue-non-SAE, R, Mild | 0.25 | 0.16 | 0.00 | 0.17 | 0.00 | 0.21
  Fatigue-non-SAE, R, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Flank Pain-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Flatulence-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Flatulence-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Folliculitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Fungal Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Furuncle-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.17 | 0.00 | 0.00 | 0.12
  Gastric Ulcer-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Gastric Ulcer-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Gastroenteritis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Gastroenteritis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Gastroenteritis-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Gastroenteritis Viral-non-SAE, NR, Mild | 0.23 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Gastroenteritis Viral-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.05 | 0.07
  Goitre-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Gravitational Oedema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Haematochezia-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Haemoglobin Decreased-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Haemorrhoids-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Head Injury-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Headache-non-SAE, NR, Mild | 0.23 | 0.17 | 0.17 | 0.08 | 0.04 | 0.08
  Headache-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.08 | 0.03 | 0.13
  Headache-non-SAE, NR, Severe | 0.00 | 0.00 | 0.17 | 0.00 | 0.07 | 0.12
  Headache-non-SAE, R, Mild | 1.10 | 0.20 | 0.17 | 0.17 | 0.11 | 0.14
  Headache-non-SAE, R, Moderate | 0.63 | 0.07 | 0.17 | 0.00 | 0.00 | 0.24
  Headache-non-SAE, R, Severe | 0.38 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Heart Rate Decreased-non-SAE, R, Mild | 0.00 | 0.00 | 0.50 | 0.00 | 0.00 | 0.50
  Heart Rate Increased-non-SAE, NR, Mild | 0.00 | 0.25 | 0.00 | 0.08 | 0.00 | 0.17
  Heart Rate Increased-non-SAE, R, Mild | 0.25 | 0.08 | 0.25 | 0.08 | 0.03 | 0.08
  Heart Rate Increased-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Hiatus Hernia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Hordeolum-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Hyperlipidaemia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Hypoxia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Implant Site Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Infection-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Infection-non-SAE, NR, Moderate | 0.20 | 0.08 | 0.17 | 0.00 | 0.04 | 0.08
  Influenza-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.03 | 0.08
  Influenza-non-SAE, NR, Moderate | 0.23 | 0.07 | 0.00 | 0.08 | 0.04 | 0.07
  Infusion Related Reaction-non-SAE, R, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Erythema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Haematoma-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.03 | 0.06
  Infusion Site Haematoma-non-SAE, R, Mild | 0.00 | 0.07 | 0.17 | 0.17 | 0.04 | 0.07
  Infusion Site Haematoma-non-SAE, R, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Infusion Site Haemorrhage-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Irritation-non-SAE, R, Mild | 0.25 | 0.10 | 0.00 | 0.00 | 0.05 | 0.07
  Infusion Site Oedema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Pain-non-SAE, R, Mild | 0.20 | 0.14 | 0.15 | 0.08 | 0.04 | 0.16
  Infusion Site Pain-non-SAE, R, Moderate | 0.00 | 0.07 | 0.17 | 0.16 | 0.00 | 0.16
  Infusion Site Pruritus-non-SAE, NR, Moderate | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Infusion Site Pruritus-non-SAE, R, Mild | 0.00 | 0.15 | 0.17 | 0.08 | 0.00 | 0.16
  Infusion Site Pruritus-non-SAE, R, Moderate | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Infusion Site Rash-non-SAE, NR, Mild | 0.00 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Infusion Site Rash-non-SAE, R, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.03 | 0.08
  Infusion Site Reaction-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Infusion Site Swelling-non-SAE, R, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Infusion Site Swelling-non-SAE, R, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Vesicles-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Inguinal Mass-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Injection Site Haematoma-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Injection Site Haematoma-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Injection Site Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Insomnia-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.03 | 0.03
  Insomnia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Intermit. Explosive Disorder-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Irritability-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.13 | 0.13
  Irritable Bowel Syndrome-non-SAE, NR, Moderate | 0.00 | 0.06 | 0.00 | 0.08 | 0.04 | 0.06
  Joint Dislocation-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Joint Sprain-non-SAE, NR, Mild | 0.00 | 0.17 | 0.00 | 0.00 | 0.00 | 0.17
  Joint Swelling-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Joint Swelling-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Laryngitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Laryngitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Laryngitis Viral-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Lethargy-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Limb Injury-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Lip Ulceration-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Livedo Reticularis-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lung Infection-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lung Infection-non-SAE, NR, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lymphadenopathy-non-SAE, NR, Mild | 0.25 | 0.00 | 0.17 | 0.00 | 0.04 | 0.05
  Malaise-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Malaise-non-SAE, R, Moderate | 0.00 | 0.10 | 0.00 | 0.00 | 0.00 | 0.10
  Memory Impairment-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Middle Ear Effusion-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Migraine-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.03 | 0.06
  Migraine-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Migraine-non-SAE, NR, Severe | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Migraine-non-SAE, R, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Migraine-non-SAE, R, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Mouth Ulceration-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Muscle Strain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.03 | 0.10
  Muscular Weakness-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Musculoskeletal Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Musculoskeletal Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.07 | 0.04 | 0.07
  Myalgia-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.08 | 0.09 | 0.09
  Myalgia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Myopia-non-SAE, NR, Mild | 0.00 | 0.10 | 0.00 | 0.00 | 0.00 | 0.10
  Nasal Congestion-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.06 | 0.06
  Nasal Congestion-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.04 | 0.10
  Nasal Disorder-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Nasal Mucosal Disorder-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Nasal Polyps-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Nasopharyngitis-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.08 | 0.04 | 0.04
  Nasopharyngitis-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.07 | 0.07 | 0.07
  Nausea-non-SAE, NR, Mild | 0.25 | 0.08 | 0.17 | 0.08 | 0.12 | 0.08
  Nausea-non-SAE, NR, Moderate | 0.00 | 0.07 | 0.00 | 0.17 | 0.03 | 0.07
  Nausea-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Nausea-non-SAE, R, Mild | 0.75 | 0.08 | 0.17 | 0.27 | 0.04 | 0.13
  Nausea-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Oedema Peripheral-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Oedema Peripheral-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Oral Herpes-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.03 | 0.07
  Oropharyngeal Pain-non-SAE, NR, Mild | 0.20 | 0.08 | 0.00 | 0.00 | 0.07 | 0.07
  Oropharyngeal Pain-non-SAE, NR, Moderate | 0.23 | 0.00 | 0.00 | 0.08 | 0.05 | 0.07
  Osteomyelitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Osteopenia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Otitis Externa-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Otitis Media-non-SAE, NR, Mild | 0.00 | 0.13 | 0.17 | 0.00 | 0.00 | 0.17
  Otitis Media-non-SAE, NR, Moderate | 0.00 | 0.17 | 0.00 | 0.13 | 0.11 | 0.14
  Pain-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Pain In Extremity-non-SAE, NR, Mild | 0.38 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Pain In Extremity-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.08 | 0.00 | 0.13
  Pain In Extremity-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Pain In Extremity-non-SAE, R, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Paraesthesia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Paronychia-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Periorbital Oedema-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Pharyngitis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.05 | 0.07
  Pharyngitis-non-SAE, NR, Moderate | 0.50 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Pharyngitis Streptococcal-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Pneumonia-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Pneumonia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.04 | 0.06
  Pneumonia Bacterial-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Pneumonia Streptococcal-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Procedural Pain-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.04 | 0.04
  Pyrexia-non-SAE, NR, Mild | 0.25 | 0.07 | 0.00 | 0.00 | 0.07 | 0.07
  Pyrexia-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Pyrexia-non-SAE, R, Mild | 0.63 | 0.17 | 0.00 | 0.00 | 0.07 | 0.07
  Pyrexia-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Rales-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rash-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rash-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Rash Erythematous-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.05 | 0.07
  Rash Macular-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rash Papular-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Rash Pruritic-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Respiratory Rate Increased-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Respir. Tract Infect. Viral-non-SAE, NR, Mild | 0.25 | 0.17 | 0.00 | 0.00 | 0.03 | 0.10
  Respir. Tract Infect Viral-non-SAE, NR, Moderate | 0.25 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Rhinitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.09 | 0.09
  Rhinitis Allergic-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rhinorrhoea-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Road Traffic Accident-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Scleritis-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Scleritis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Scoliosis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Sinus Congestion-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Sinus Congestion-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Sinus Disorder-non-SAE, NR, Severe | 0.00 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Sinus Headache-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Sinus Headache-non-SAE, NR, Moderate | 0.50 | 0.07 | 0.00 | 0.08 | 0.00 | 0.08
  Sinusitis-non-SAE, NR, Mild | 0.46 | 0.00 | 0.00 | 0.08 | 0.04 | 0.04
  Sinusitis-non-SAE, NR, Moderate | 0.25 | 0.07 | 0.17 | 0.08 | 0.04 | 0.08
  Sinusitis-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Sinusitis Fungal-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Skin Laceration-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Skin Lesion-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Skin Papilloma-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Skin Warm-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Sports Injury-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Streptococcal Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Subcutaneous Abscess-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Suicidal Ideation-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Sunburn-non-SAE, NR, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Tendonitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Tooth Fracture-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Tooth Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Toothache-non-SAE, NR, Moderate | 0.00 | 0.07 | 0.00 | 0.00 | 0.03 | 0.05
  Tourette's Disorder-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Upper Respir. Tract Congestion-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Upper Respir. Tract Infection-non-SAE, NR, Mild | 0.25 | 0.08 | 0.17 | 0.08 | 0.05 | 0.08
  Upper Respir. Tract Infect.-non-SAE, NR, Moderate | 0.25 | 0.08 | 0.00 | 0.08 | 0.05 | 0.07
  Urinary Tract Infection-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Urticaria-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Urticaria-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Vaginal Lesion-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Vaginitis Bacterial-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Varicose Vein-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Varicose Vein-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Vestibulitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Viral Infection-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Viral Infection-non-SAE, NR, Moderate | 0.38 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Viral Skin Infection-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Viral Upper Respir. Tract Infect-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Viral Up. Respir Tract Infec-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Vitamin D Deficiency-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Vomiting-non-SAE, NR, Mild | 0.25 | 0.07 | 0.17 | 0.08 | 0.04 | 0.07
  Vomiting-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Vomiting-non-SAE, R, Mild | 0.75 | 0.00 | 0.00 | 0.09 | 0.05 | 0.07
  Vomiting-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.18 | 0.00 | 0.18
  Vulvovaginal Candidiasis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Vulvovaginal Mycotic Infection-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Vulvovaginal Mycotic Infect.-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Wheezing-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.09 | 0.09
  Wound-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08

31. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Severity, and Causality (SNSC -All Ages)
Description: as for outcome 29
Time Frame: Throughout entire study (1 year and 9 months)
Population: Study participants who are naïve to SC administration of immunoglobulins and received any study drug during each of the study parts
Measure: Number; unit: Adverse events
Arm/Group | Study Part 1, IV Administration | Study Part 2, SC Administration | Study Part 3a, SC Administration | Study Part 3b, SC Administration | Study Extension, SC Administration | Total SC (Study Parts 2, 3a, 3b, Extension)
Number analyzed (Participants) | 38 | 36 | 34 | 34 | 27 | 36
Adverse events
  Abdominal Discomfort- non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Abdominal Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Abdominal Pain-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Abdominal Pain Upper-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 2 | 2
  Abdominal Pain Upper-non-SAE, R, Mild | 0 | 3 | 0 | 0 | 0 | 3
  Acne-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Acute Sinusitis-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Alopecia-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Ammonia Increased-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Animal Bite-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Anorexia-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Anxiety-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Aphthous Stomatitis-non-SAE, NR, Mild | 0 | 1 | 1 | 0 | 2 | 4
  Arthralgia-non-SAE, NR, Moderate | 0 | 2 | 0 | 0 | 0 | 2
  Arthralgia-non-SAE, R, Mild | 1 | 0 | 1 | 0 | 0 | 1
  Arthralgia-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Arthritis-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Arthropod Bite-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 1 | 2
  Asthenia-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Asthma-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Asthma-non-SAE, NR, Moderate | 3 | 0 | 1 | 1 | 3 | 5
  Asthma-non-SAE, NR, Severe | 0 | 0 | 0 | 1 | 0 | 1
  Asthma-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Asthma Exercise Induced-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  ADHD-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Back Pain-non-SAE, NR, Mild | 1 | 0 | 0 | 1 | 0 | 1
  Back Pain-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Back Pain-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Biliary Tract Infection Bacterial-SAE, NR, Moderat | 0 | 1 | 0 | 0 | 0 | 1
  Blepharitis-non-SAE,NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  B.P. Diastolic Decreased-non-SAE, R, Mild | 0 | 0 | 2 | 0 | 0 | 2
  Blood Pressure Increased-non-SAE, NR, Mild | 0 | 0 | 0 | 2 | 0 | 2
  Blood Pressure Increased-non-SAE, R, Mild | 0 | 0 | 0 | 1 | 0 | 1
  B.P. Systolic Increased-non-SAE, NR, Mild | 0 | 1 | 1 | 0 | 0 | 2
  B.P. Systolic Increased-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  B.P. Systolic Increased-non-SAE, R, Mild | 1 | 4 | 2 | 0 | 0 | 6
  B.P. Systolic Increased-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Breast Tenderness-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Bronchitis-non-SAE, NR, Mild | 1 | 1 | 0 | 2 | 2 | 5
  Bronchitis-non-SAE, NR, Moderate | 1 | 0 | 1 | 0 | 2 | 3
  Bursitis-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Candidiasis-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Cardiac Murmur-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Centrl Venous Catheterisation-non-SAE, NR, Moderat | 0 | 0 | 0 | 0 | 1 | 1
  Cervical Spinal Stenosis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Chest Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Chest Pain-SAE, NR, Severe | 0 | 0 | 0 | 1 | 0 | 1
  Chills-non-SAE, R, Mild | 7 | 0 | 0 | 0 | 0 | 0
  Chills-non-SAE, R, Moderate | 6 | 0 | 0 | 0 | 0 | 0
  C.O.P.D.-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  C.O.P.D.-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Chronic Sinusitis-non-SAE, NR, Mild | 0 | 0 | 1 | 1 | 1 | 3
  Confusional State-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Conjunctival Hyperaemia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Conjunctivitis Allergic-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Conjunctivitis Infective-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Constipation-non-SAE, NR, Mild | 1 | 2 | 0 | 0 | 1 | 3
  Constipation-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Contusion-non-SAE, NR, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Contusion-non-SAE, R, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Convulsion-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Convulsion-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Cough-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Cough-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Croup Infectious-non-SAE, NR, Mild | 0 | 2 | 0 | 1 | 0 | 3
  Croup Infectious-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Cryptosporidiosis Infection-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Dental Caries-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Dermatitis-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Dermatitis Contact-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Device Failure-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Diarrhoea-non-SAE, NR, Mild | 1 | 1 | 0 | 0 | 1 | 2
  Diarrhoea-non-SAE, NR, Moderate | 1 | 2 | 1 | 0 | 0 | 3
  Diarrhoea-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 1 | 1
  Diarrhoea Haemorrhagic-non-SAE, NR,Mild | 1 | 0 | 0 | 0 | 0 | 0
  Diarrhoea Infectious-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Diverticulitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Drug Eruption-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dyspnoea-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Dyspnoea-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Ear Infection-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 1 | 1
  Ear Pain-non-SAE, NR, Mild | 0 | 1 | 1 | 0 | 1 | 3
  Ear Pain-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Eczema-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 3 | 4
  Eczema-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Epistaxis-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Epistaxis-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 1 | 2
  Excoriation-non-SAE, NR, Mild | 0 | 0 | 0 | 2 | 0 | 2
  Eye Infection Viral-non-SAE, NR, Moderate | 3 | 1 | 0 | 1 | 1 | 3
  Fall-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Fatigue-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Fatigue-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Fatigue-non-SAE, R, Mild | 1 | 3 | 0 | 2 | 0 | 5
  Fatigue-non-SAE, R, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Flank Pain-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Fungal Infection-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Furuncle-non-SAE, NR, Moderate | 0 | 1 | 1 | 0 | 0 | 2
  Gastric Ulcer-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Gastric Ulcer-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Gastroenteritis-non-SAE, NR, Mild | 1 | 0 | 0 | 1 | 0 | 1
  Gastroenteritis-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Gastroenteritis-non-SAE, R, Mild | 0 | 2 | 0 | 0 | 0 | 0
  Gastroenteritis Viral-non-SAE, NR, Mild | 1 | 2 | 0 | 0 | 0 | 2
  Gastroenteritis Viral-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 3 | 4
  Goitre-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Gravitational Oedema-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Haematochezia-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Haemoglobin Decreased-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Haemorrhoids-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Head Injury-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Headache-non-SAE, NR, Mild | 7 | 3 | 2 | 3 | 8 | 16
  Headache-non-SAE, NR, Moderate | 4 | 0 | 2 | 1 | 1 | 4
  Headache-non-SAE, NR, Severe | 0 | 0 | 1 | 0 | 1 | 2
  Headache-non-SAE, R, Mild | 19 | 4 | 1 | 2 | 8 | 15
  Headache-non-SAE, R, Moderate | 8 | 1 | 1 | 0 | 0 | 2
  Headache-non-SAE, R, Severe | 3 | 1 | 0 | 0 | 0 | 1
  Heart Rate Decreased-non-SAE, R, Mild | 0 | 0 | 3 | 0 | 0 | 3
  Heart Rate Increased-non-SAE, NR, Mild | 0 | 3 | 0 | 1 | 0 | 4
  Heart Rate Increased-non-SAE, R, Mild | 4 | 4 | 3 | 1 | 1 | 9
  Heart Rate Increased-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Hiatus Hernia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Hordeolum-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Hyperlipidaemia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Hypoxia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Implant Site Pain-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Infection-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 1 | 1
  Infection-non-SAE, NR, Moderate | 1 | 1 | 0 | 0 | 0 | 1
  Influenza-non-SAE, NR, Mild | 1 | 3 | 0 | 0 | 2 | 5
  Influenza-non-SAE, NR, Moderate | 1 | 4 | 0 | 0 | 2 | 6
  Infusion Related Reaction-non-SAE, R, Mild | 1 | 1 | 0 | 0 | 0 | 1
  Infusion Site Erythema-non-SAE, R, Mild | 0 | 3 | 0 | 0 | 0 | 3
  Infusion Site Haematoma-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 1 | 2
  Infusion Site Haematoma-non-SAE, R, Mild | 0 | 2 | 2 | 2 | 5 | 11
  Infusion Site Haematoma-non-SAE, R, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Infusion Site Haemorrhage-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Irritation-non-SAE, R, Mild | 1 | 1 | 0 | 0 | 0 | 1
  Infusion Site Oedema-non-SAE, R, Mild | 0 | 2 | 0 | 0 | 0 | 2
  Infusion Site Pain-non-SAE, R, Mild | 1 | 8 | 2 | 2 | 1 | 13
  Infusion Site Pain-non-SAE, R, Moderate | 0 | 5 | 1 | 2 | 0 | 8
  Infusion Site Pruritus-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Pruritus-non-SAE, R, Mild | 0 | 1 | 1 | 1 | 0 | 3
  Infusion Site Pruritus-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Rash-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Rash-non-SAE, R, Mild | 0 | 1 | 1 | 0 | 1 | 3
  Infusion Site Reaction-non-SAE, R, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Infusion Site Swelling-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Swelling-non-SAE, R, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Infusion Site Vesicles-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Inguinal Mass-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Injection Site Haematoma-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Insomnia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 2 | 3
  Insomnia-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Intermit. Explosive Disorder-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Irritability-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Irritable Bowel Syndrome-non-SAE, NR, Moderate | 0 | 1 | 0 | 1 | 1 | 3
  Joint Dislocation-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Laryngitis-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Laryngitis-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Lethargy-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Limb Injury-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Lip Ulceration-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Livedo Reticularis-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Lung Infection-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Lung Infection-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Lymphadenopathy-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 2 | 2
  Malaise-non-SAE, NR, Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Malaise-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Middle Ear Effusion-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Migraine-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 1 | 2
  Migraine-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Migraine-non-SAE, R, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Mouth Ulceration-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Muscular Weakness-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Musculoskeletal Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Musculoskeletal Pain-non-SAE, NR, Moderate | 0 | 0 | 1 | 1 | 1 | 3
  Myalgia-non-SAE, NR, Mild | 0 | 1 | 1 | 1 | 5 | 8
  Myalgia-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Myopia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Nasal Congestion-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Nasal Congestion-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Nasal Disorder-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Nasal Mucosal Disorder-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Nasal Polyps-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Nasopharyngitis-non-SAE, NR, Mild | 3 | 0 | 0 | 1 | 2 | 3
  Nasopharyngitis-non-SAE, NR, Moderate | 0 | 1 | 0 | 1 | 2 | 4
  Nausea-non-SAE, NR, Mild | 1 | 2 | 0 | 1 | 1 | 4
  Nausea-non-SAE, NR, Moderate | 0 | 1 | 0 | 2 | 1 | 4
  Nausea-non-SAE, NR, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Nausea-non-SAE, R, Mild | 4 | 0 | 0 | 3 | 0 | 3
  Oedema Peripheral-non-SAE, R, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Oral Herpes-non-SAE, NR, Mild | 0 | 2 | 0 | 0 | 1 | 3
  Oropharyngeal Pain-non-SAE, NR, Mild | 0 | 2 | 0 | 0 | 3 | 5
  Oropharyngeal Pain-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 1 | 2
  Osteomyelitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Otitis Externa-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Otitis Media-non-SAE, NR, Mild | 0 | 3 | 1 | 0 | 0 | 4
  Otitis Media-non-SAE, NR, Moderate | 0 | 2 | 0 | 3 | 2 | 7
  Pain-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Pain In Extremity-non-SAE, NR, Mild | 3 | 0 | 0 | 0 | 0 | 0
  Pain In Extremity-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Pain In Extremity-non-SAE, R, Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Pain In Extremity-non-SAE, R, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Paraesthesia-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Paronychia-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Periorbital Oedema-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Pharyngitis-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Pharyngitis-non-SAE, NR, Moderate | 2 | 1 | 0 | 1 | 0 | 2
  Pharyngitis Streptococcal-non-SAE, NR, Moderate | 0 | 2 | 0 | 0 | 0 | 2
  Pneumonia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 2 | 3
  Pneumonia Streptococcal-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Procedural Pain-non-SAE, NR, Moderate | 1 | 0 | 0 | 1 | 2 | 3
  Pyrexia-non-SAE, NR, Mild | 1 | 2 | 0 | 0 | 9 | 11
  Pyrexia-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 2 | 2
  Pyrexia-non-SAE, R, Mild | 5 | 2 | 0 | 0 | 4 | 6
  Pyrexia-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 1 | 1
  Rash-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Rash-non-SAE, R, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Rash Erythematous-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 1 | 2
  Rash Macular-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Rash Papular-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Rash Pruritic-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Respiratory Rate Increased-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Respir. Tract Infect. Viral-non-SAE, NR, Mild | 2 | 2 | 0 | 0 | 0 | 2
  Respir. Tract Infect Viral-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Rhinitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Rhinitis Allergic-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Rhinorrhoea-non-SAE, NR, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Road Traffic Accident-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Scleritis-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Scleritis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Scoliosis-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Sinus Congestion-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 1 | 1
  Sinus Congestion-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Sinus Disorder-non-SAE, NR, Severe | 0 | 1 | 0 | 0 | 0 | 1
  Sinus Headache-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 1 | 1
  Sinus Headache-non-SAE, NR, Moderate | 2 | 1 | 0 | 1 | 0 | 2
  Sinusitis-non-SAE, NR, Mild | 3 | 0 | 0 | 1 | 3 | 4
  Sinusitis-non-SAE, NR, Moderate | 6 | 4 | 4 | 4 | 3 | 15
  Sinusitis-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Sinusitis Fungal-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Skin Laceration-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Skin Lesion-non-SAE, NR, Mild | 1 | 0 | 0 | 1 | 0 | 1
  Skin Papilloma-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Skin Warm-non-SAE, R, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Streptococcal Infection-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Subcutaneous Abscess-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Suicidal Ideation-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Sunburn-non-SAE, NR, Severe | 1 | 0 | 0 | 0 | 0 | 0
  Tendonitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Tooth Fracture-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Tooth Infection-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Toothache-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 1 | 2
  Tourette's Disorder-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Upper Respir. Tract Congestion-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Upper Respir. Tract Infection-non-SAE, NR, Mild | 2 | 3 | 3 | 5 | 7 | 18
  Upper Respir. Tract Infect.-non-SAE, NR, Moderate | 1 | 1 | 0 | 1 | 3 | 5
  Urinary Tract Infection-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Urticaria-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 2 | 2
  Urticaria-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Vaginal Lesion-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Vaginitis Bacterial-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Varicose Vein-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Varicose Vein-non-SAE, NR, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Viral Infection-non-SAE, NR, Mild | 2 | 2 | 0 | 0 | 0 | 2
  Viral Infection-non-SAE, NR, Moderate | 3 | 0 | 0 | 1 | 0 | 1
  Viral Skin Infection-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Viral Upper Respir. Tract Infect-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Vitamin D Deficiency-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Vomiting-non-SAE, NR, Mild | 1 | 1 | 1 | 1 | 4 | 7
  Vomiting-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Vomiting-non-SAE, R, Mild | 8 | 0 | 0 | 1 | 1 | 2
  Vomiting-non-SAE, R, Moderate | 1 | 0 | 0 | 2 | 0 | 2
  Vulvovaginal Candidiasis-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Vulvovaginal Mycotic Infection-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Wheezing-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1

32. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Severity, and Causality (SNSC- All Ages)
Description: as for outcome 30
Time Frame: Throughout entire study (1 year and 9 months)
Population: as for outcome 31
Measure: Number; unit: AEs per infusion
Arm/Group | Study Part 1, IV Administration | Study Part 2, SC Administration | Study Part 3a, SC Administration | Study Part 3b, SC Administration | Study Extension, SC Administration | Total SC (Parts 2, 3a, 3b, Extension)
Number analyzed (Participants) | 38 | 36 | 34 | 34 | 27 | 36
AEs per infusion
  Abdominal Discomfort- non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Abdominal Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Abdominal Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Abdominal Pain Upper-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Abdominal Pain Upper-non-SAE, R, Mild | 0.00 | 0.10 | 0.00 | 0.00 | 0.00 | 0.10
  Acne-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Acute Sinusitis-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Alopecia-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Ammonia Increased-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Animal Bite-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Anorexia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Anxiety-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Aphthous Stomatitis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.14 | 0.14
  Arthralgia-non-SAE, NR, Moderate | 0.00 | 0.11 | 0.00 | 0.00 | 0.00 | 0.11
  Arthralgia-non-SAE, R, Mild | 0.25 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Arthralgia-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Arthritis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Arthropod Bite-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.03 | 0.06
  Asthenia-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Asthma-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Asthma-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.08 | 0.03 | 0.04
  Asthma-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Asthma-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Asthma Exercise Induced-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  ADHD-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Back Pain-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Back Pain-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Back Pain-non-SAE, R, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Biliary Tract Infection Bacterial-SAE, NR, Moderat | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Blepharitis-non-SAE,NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  B.P. Diastolic Decreased-non-SAE, R, Mild | 0.00 | 0.00 | 0.33 | 0.00 | 0.00 | 0.33
  Blood Pressure Increased-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.17 | 0.00 | 0.17
  Blood Pressure Increased-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  B.P. Systolic Increased-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.00 | 0.12
  B.P. Systolic Increased-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  B.P. Systolic Increased-non-SAE, R, Mild | 0.25 | 0.16 | 0.17 | 0.00 | 0.00 | 0.17
  B.P. Systolic Increased-non-SAE, R, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Breast Tenderness-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Bronchitis-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.17 | 0.06 | 0.08
  Bronchitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.00 | 0.08 | 0.12
  Bursitis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Candidiasis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Cardiac Murmur-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Centrl Venous Catheterisation-non-SAE, NR, Moderat | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Cervical Spinal Stenosis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Chest Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Chest Pain-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Chills-non-SAE, R, Mild | 0.75 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Chills-non-SAE, R, Moderate | 0.50 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  C.O.P.D.-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  C.O.P.D.-non-SAE, NR, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Chronic Sinusitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.08 | 0.03 | 0.08
  Confusional State-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Conjunctival Hyperaemia-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Conjunctivitis Allergic-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Conjunctivitis Infective-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Constipation-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.03 | 0.07
  Constipation-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Contusion-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Contusion-non-SAE, R, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Convulsion-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Convulsion-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Cough-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Cough-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Croup Infectious-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Croup Infectious-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.11 | 0.11
  Cryptosporidiosis Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Dental Caries-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Dermatitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Dermatitis Contact-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Device Failure-non-SAE, NR, Mild | 0.23 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Diarrhoea-non-SAE, NR, Mild | 0.25 | 0.06 | 0.00 | 0.00 | 0.05 | 0.06
  Diarrhoea-non-SAE, NR, Moderate | 0.25 | 0.17 | 0.17 | 0.00 | 0.00 | 0.17
  Diarrhoea-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Diarrhoea Haemorrhagic-non-SAE, NR,Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Diarrhoea Infectious-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Diverticulitis-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Drug Eruption-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Dyspnoea-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Dyspnoea-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Ear Infection-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Ear Pain-non-SAE, NR, Mild | 0.00 | 0.06 | 0.17 | 0.00 | 0.03 | 0.06
  Ear Pain-non-SAE, R, Moderate | 0.00 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Eczema-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.04 | 0.06
  Eczema-non-SAE, NR, Severe | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Epistaxis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Epistaxis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.14 | 0.00 | 0.07 | 0.10
  Excoriation-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.17 | 0.00 | 0.17
  Eye Infection Viral-non-SAE, NR, Moderate | 0.38 | 0.10 | 0.00 | 0.08 | 0.04 | 0.08
  Fall-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Fatigue-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.11 | 0.11
  Fatigue-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Fatigue-non-SAE, R, Mild | 0.25 | 0.17 | 0.00 | 0.17 | 0.00 | 0.22
  Fatigue-non-SAE, R, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Flank Pain-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Fungal Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Furuncle-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.17 | 0.00 | 0.00 | 0.12
  Gastric Ulcer-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Gastric Ulcer-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Gastroenteritis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Gastroenteritis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Gastroenteritis-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Gastroenteritis Viral-non-SAE, NR, Mild | 0.20 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Gastroenteritis Viral-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.05 | 0.07
  Goitre-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Gravitational Oedema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Haematochezia-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Haemoglobin Decreased-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Haemorrhoids-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Head Injury-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Headache-non-SAE, NR, Mild | 0.25 | 0.13 | 0.17 | 0.08 | 0.04 | 0.07
  Headache-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.08 | 0.03 | 0.13
  Headache-non-SAE, NR, Severe | 0.00 | 0.00 | 0.17 | 0.00 | 0.07 | 0.12
  Headache-non-SAE, R, Mild | 1.10 | 0.23 | 0.17 | 0.17 | 0.11 | 0.18
  Headache-non-SAE, R, Moderate | 0.63 | 0.07 | 0.17 | 0.00 | 0.00 | 0.24
  Headache-non-SAE, R, Severe | 0.38 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Heart Rate Decreased-non-SAE, R, Mild | 0.00 | 0.00 | 0.50 | 0.00 | 0.00 | 0.50
  Heart Rate Increased-non-SAE, NR, Mild | 0.00 | 0.25 | 0.00 | 0.08 | 0.00 | 0.17
  Heart Rate Increased-non-SAE, R, Mild | 0.25 | 0.08 | 0.25 | 0.08 | 0.03 | 0.08
  Heart Rate Increased-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Hiatus Hernia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Hordeolum-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Hyperlipidaemia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Hypoxia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Implant Site Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Infection-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Infection-non-SAE, NR, Moderate | 0.20 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Influenza-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.03 | 0.08
  Influenza-non-SAE, NR, Moderate | 0.20 | 0.07 | 0.00 | 0.00 | 0.04 | 0.06
  Infusion Related Reaction-non-SAE, R, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Erythema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Haematoma-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.03 | 0.06
  Infusion Site Haematoma-non-SAE, R, Mild | 0.00 | 0.07 | 0.17 | 0.17 | 0.04 | 0.08
  Infusion Site Haematoma-non-SAE, R, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Infusion Site Haemorrhage-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Irritation-non-SAE, R, Mild | 0.25 | 0.10 | 0.00 | 0.00 | 0.05 | 0.07
  Infusion Site Oedema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Pain-non-SAE, R, Mild | 0.20 | 0.14 | 0.15 | 0.08 | 0.04 | 0.16
  Infusion Site Pain-non-SAE, R, Moderate | 0.00 | 0.07 | 0.17 | 0.16 | 0.00 | 0.16
  Infusion Site Pruritus-non-SAE, NR, Moderate | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Infusion Site Pruritus-non-SAE, R, Mild | 0.00 | 0.07 | 0.17 | 0.08 | 0.00 | 0.08
  Infusion Site Pruritus-non-SAE, R, Moderate | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Infusion Site Rash-non-SAE, NR, Mild | 0.00 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Infusion Site Rash-non-SAE, R, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.03 | 0.08
  Infusion Site Reaction-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Infusion Site Swelling-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Swelling-non-SAE, R, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Infusion Site Vesicles-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Inguinal Mass-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Injection Site Haematoma-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Insomnia-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.03 | 0.03
  Insomnia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Intermit. Explosive Disorder-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Irritability-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.13 | 0.13
  Irritable Bowel Syndrome-non-SAE, NR, Moderate | 0.00 | 0.06 | 0.00 | 0.08 | 0.04 | 0.06
  Joint Dislocation-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Laryngitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Laryngitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Lethargy-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Limb Injury-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Lip Ulceration-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Livedo Reticularis-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lung Infection-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lung Infection-non-SAE, NR, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lymphadenopathy-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Malaise-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Malaise-non-SAE, R, Moderate | 0.00 | 0.10 | 0.00 | 0.00 | 0.00 | 0.10
  Middle Ear Effusion-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Migraine-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.03 | 0.06
  Migraine-non-SAE, NR, Severe | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Migraine-non-SAE, R, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Mouth Ulceration-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Muscular Weakness-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.09 | 0.00 | 0.09
  Musculoskeletal Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Musculoskeletal Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.07 | 0.04 | 0.07
  Myalgia-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.08 | 0.09 | 0.9
  Myalgia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Myopia-non-SAE, NR, Mild | 0.00 | 0.10 | 0.00 | 0.00 | 0.00 | 0.10
  Nasal Congestion-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Nasal Congestion-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Nasal Disorder-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Nasal Mucosal Disorder-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Nasal Polyps-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Nasopharyngitis-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.04 | 0.05
  Nasopharyngitis-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.07 | 0.06 | 0.07
  Nausea-non-SAE, NR, Mild | 0.25 | 0.07 | 0.00 | 0.08 | 0.07 | 0.08
  Nausea-non-SAE, NR, Moderate | 0.00 | 0.07 | 0.00 | 0.17 | 0.03 | 0.07
  Nausea-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Nausea-non-SAE, R, Mild | 0.75 | 0.00 | 0.00 | 0.27 | 0.00 | 0.27
  Oedema Peripheral-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Oral Herpes-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.03 | 0.07
  Oropharyngeal Pain-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.07 | 0.07
  Oropharyngeal Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.07 | 0.08
  Osteomyelitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Otitis Externa-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Otitis Media-non-SAE, NR, Mild | 0.00 | 0.13 | 0.17 | 0.00 | 0.00 | 0.17
  Otitis Media-non-SAE, NR, Moderate | 0.00 | 0.17 | 0.00 | 0.13 | 0.11 | 0.14
  Pain-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Pain In Extremity-non-SAE, NR, Mild | 0.38 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Pain In Extremity-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Pain In Extremity-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Pain In Extremity-non-SAE, R, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Paraesthesia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Paronychia-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Periorbital Oedema-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Pharyngitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Pharyngitis-non-SAE, NR, Moderate | 0.50 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Pharyngitis Streptococcal-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Pneumonia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.04 | 0.06
  Pneumonia Streptococcal-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Procedural Pain-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.04 | 0.04
  Pyrexia-non-SAE, NR, Mild | 0.25 | 0.06 | 0.00 | 0.00 | 0.12 | 0.07
  Pyrexia-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Pyrexia-non-SAE, R, Mild | 0.63 | 0.17 | 0.00 | 0.00 | 0.07 | 0.07
  Pyrexia-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Rash-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rash-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Rash Erythematous-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.05 | 0.07
  Rash Macular-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rash Papular-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Rash Pruritic-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Respiratory Rate Increased-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Respir. Tract Infect. Viral-non-SAE, NR, Mild | 0.25 | 0.17 | 0.00 | 0.00 | 0.00 | 0.17
  Respir. Tract Infect Viral-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Rhinitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.09 | 0.09
  Rhinitis Allergic-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Rhinorrhoea-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Road Traffic Accident-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Scleritis-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Scleritis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Scoliosis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Sinus Congestion-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Sinus Congestion-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Sinus Disorder-non-SAE, NR, Severe | 0.00 | 0.06 | 0.00 | 0.00 | 0.00 | 0.06
  Sinus Headache-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Sinus Headache-non-SAE, NR, Moderate | 0.50 | 0.07 | 0.00 | 0.08 | 0.00 | 0.08
  Sinusitis-non-SAE, NR, Mild | 0.46 | 0.00 | 0.00 | 0.08 | 0.04 | 0.04
  Sinusitis-non-SAE, NR, Moderate | 0.25 | 0.07 | 0.17 | 0.08 | 0.04 | 0.08
  Sinusitis-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Sinusitis Fungal-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Skin Laceration-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Skin Lesion-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Skin Papilloma-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Skin Warm-non-SAE, R, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Streptococcal Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Subcutaneous Abscess-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Suicidal Ideation-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Sunburn-non-SAE, NR, Severe | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Tendonitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Tooth Fracture-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Tooth Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Toothache-non-SAE, NR, Moderate | 0.00 | 0.07 | 0.00 | 0.00 | 0.03 | 0.05
  Tourette's Disorder-non-SAE, NR, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Upper Respir. Tract Congestion-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Upper Respir. Tract Infection-non-SAE, NR, Mild | 0.23 | 0.08 | 0.17 | 0.08 | 0.06 | 0.08
  Upper Respir. Tract Infect.-non-SAE, NR, Moderate | 0.25 | 0.08 | 0.00 | 0.08 | 0.05 | 0.07
  Urinary Tract Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Urticaria-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.05 | 0.05
  Urticaria-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Vaginal Lesion-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Vaginitis Bacterial-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Varicose Vein-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Varicose Vein-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Viral Infection-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Viral Infection-non-SAE, NR, Moderate | 0.38 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Viral Skin Infection-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Viral Upper Respir. Tract Infect-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Vitamin D Deficiency-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Vomiting-non-SAE, NR, Mild | 0.25 | 0.07 | 0.17 | 0.08 | 0.04 | 0.07
  Vomiting-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Vomiting-non-SAE, R, Mild | 0.75 | 0.00 | 0.00 | 0.09 | 0.05 | 0.07
  Vomiting-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.18 | 0.00 | 0.18
  Vulvovaginal Candidiasis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Vulvovaginal Mycotic Infection-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Wheezing-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.09 | 0.09

33. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Severity, and Causality (SESC)
Description: as for outcome 29
Time Frame: Throughout entire study (1 year and 9 months)
Population: All study participants with prior experience with subcutaneous administration of immunoglobulins who received any study drug during each of the study parts
Measure: Number; unit: Adverse events
Arm/Group | Study Part 1, IV Administration | Study Part 2, SC Administration | Study Part 3a, SC Administration | Study Part 3b, SC Administration | Study Extension, SC Administration | Total SC (Parts 2, 3a, 3b, Extension)
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 11
Adverse events
  Abdominal Discomfort- non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Abdominal Distension-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 7 | 7
  Abdominal Distension-non-SAE, NR, Moderate | 0 | 0 | 0 | 2 | 2 | 4
  Abdominal Distension-non-SAE, R, Mild | 0 | 1 | 0 | 1 | 0 | 2
  Abdominal Distension-non-SAE, R, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Abdominal Pain-non-SAE, NR, Mild | 1 | 0 | 1 | 0 | 0 | 1
  Abdominal Pain Upper-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 4 | 4
  Abdominal Pain Upper-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Abdominal Pain Upper-non-SAE, R, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Abdominal Tenderness-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Acne-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Addison's Disease-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Addison's Disease-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Arthralgia-non-SAE, NR, Moderate | 0 | 1 | 1 | 2 | 1 | 5
  Arthralgia-non-SAE, NR, Severe | 0 | 0 | 0 | 0 | 1 | 1
  Asthenia-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Back Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Back Pain-non-SAE, NR, Moderate | 0 | 0 | 0 | 2 | 0 | 2
  Blepharitis-non-SAE,NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Breath Sounds Abnormal-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Bronchitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Chronic Sinusitis-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Chronic Sinusitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Conjunctivitis Bacterial-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Conjunctivitis Infective-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Costochondritis-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Costochondritis-non-SAE, NR, Severe | 0 | 1 | 0 | 0 | 0 | 1
  Cough-non-SAE, NR, Mild | 2 | 0 | 0 | 0 | 0 | 0
  Cystitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Dermatitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dermatitis Contact-non-SAE, NR, Moderate | 1 | 1 | 0 | 1 | 0 | 2
  Diarrhoea-non-SAE, NR, Mild | 0 | 1 | 0 | 2 | 1 | 4
  Diarrhoea-non-SAE, NR, Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Diarrhoea-non-SAE, R, Mild | 0 | 0 | 2 | 0 | 0 | 2
  Dyspepsia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Dyspnoea-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 0 | 1
  Ear Pain-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 1 | 1
  Exostosis-non-SAE, NR,Mild | 0 | 0 | 1 | 0 | 0 | 1
  Eye Infection Viral-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Eye Irritation-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Eye Oedema-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Fatigue-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Flatulence-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Flatulence-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Folliculitis-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Gastroenteritis Viral-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Headache-non-SAE, NR, Mild | 1 | 2 | 1 | 1 | 0 | 4
  Headache-non-SAE, R, Mild | 0 | 2 | 0 | 0 | 0 | 2
  Infection-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 1 | 2
  Influenza-non-SAE, NR, Moderate | 1 | 0 | 0 | 1 | 0 | 1
  Infusion Site Haematoma-non-SAE, R, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Infusion Site Haemorrhage-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Oedema-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Pain-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Infusion Site Pruritus-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Injection Site Haematoma-non-SAE, R, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Injection Site Pain-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Joint Sprain-non-SAE, NR, Mild | 0 | 2 | 0 | 0 | 0 | 2
  Joint Swelling-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Joint Swelling-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Laryngitis Viral-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Limb Injury-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Lymphadenopathy-non-SAE, NR, Mild | 1 | 0 | 1 | 0 | 0 | 1
  Memory Impairment-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Migraine-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Migraine-non-SAE, R, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Muscle Strain-non-SAE, NR, Mild | 0 | 0 | 1 | 0 | 1 | 2
  Nasal Congestion-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Nasal Congestion-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Nasopharyngitis-non-SAE, NR, Mild | 2 | 1 | 0 | 0 | 2 | 3
  Nasopharyngitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Nausea-non-SAE, NR, Mild | 0 | 1 | 1 | 1 | 4 | 7
  Nausea-non-SAE, R, Mild | 0 | 1 | 1 | 0 | 1 | 3
  Nausea-non-SAE, R, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Oedema Peripheral-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Oral Herpes-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Oropharyngeal Pain-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Oropharyngeal Pain-non-SAE, NR, Moderate | 2 | 0 | 0 | 0 | 1 | 1
  Osteopenia-non-SAE, NR, Moderate | 0 | 1 | 0 | 0 | 0 | 1
  Pain In Extremity-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 0 | 1
  Pharyngitis-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Pharyngitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Pneumonia-non-SAE, NR, Mild | 0 | 0 | 0 | 1 | 0 | 1
  Pneumonia Bacterial-non-SAE, NR, Moderate | 0 | 0 | 1 | 0 | 0 | 1
  Pyrexia-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 1 | 2
  Rales-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Respir. Tract Infect. Viral-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Respir. Tract Infect Viral-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Sinusitis-non-SAE, NR, Mild | 0 | 0 | 0 | 0 | 1 | 1
  Sinusitis-non-SAE, NR, Moderate | 1 | 0 | 2 | 1 | 0 | 3
  Sports Injury-non-SAE, NR, Mild | 0 | 1 | 0 | 0 | 0 | 1
  Upper Respir. Tract Infection-non-SAE, NR, Mild | 2 | 0 | 0 | 1 | 1 | 2
  Upper Respir. Tract Infect.-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Urinary Tract Infection-non-SAE, NR, Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Vestibulitis-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Viral Up. Respir Tract Infec-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Vomiting-non-SAE, NR, Mild | 1 | 0 | 0 | 0 | 0 | 0
  Vulvovaginal Mycotic Infect.-non-SAE, NR, Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Wound-non-SAE, NR, Moderate | 0 | 0 | 0 | 1 | 0 | 1

34. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Severity, and Causality (SESC)
Description: as for outcome 30
Time Frame: Throughout entire study (1 year and 9 months)
Population: as for outcome 33
Measure: Number; unit: AEs per infusion
Arm/Group | Study Part 1, IV Administration | Study Part 2, SC Administration | Study Part 3a, SC Administration | Study Part 3b, SC Administration | Study Extension, SC Administration | Total SC (Parts 2, 3a, 3b, Extension)
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 11
AEs per infusion
  Abdominal Discomfort- non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Abdominal Distension-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.29 | 0.29
  Abdominal Distension-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.17 | 0.08 | 0.13
  Abdominal Distension-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Abdominal Distension-non-SAE, R, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Abdominal Pain-non-SAE, NR, Mild | 0.25 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Abdominal Pain Upper-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.17 | 0.17
  Abdominal Pain Upper-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.08 | 0.08
  Abdominal Pain Upper-non-SAE, R, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Abdominal Tenderness-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Acne-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Addison's Disease-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Addison's Disease-non-SAE, NR, Moderate | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Arthralgia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.17 | 0.17 | 0.04 | 0.13
  Arthralgia-non-SAE, NR, Severe | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Asthenia-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Back Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Back Pain-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.17 | 0.00 | 0.17
  Blepharitis-non-SAE,NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Breath Sounds Abnormal-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Bronchitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Chronic Sinusitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Chronic Sinusitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Conjunctivitis Bacterial-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Conjunctivitis Infective-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Costochondritis-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Costochondritis-non-SAE, NR, Severe | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Cough-non-SAE, NR, Mild | 0.50 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Cystitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Dermatitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Dermatitis Contact-non-SAE, NR, Moderate | 0.25 | 0.08 | 0.00 | 0.08 | 0.00 | 0.08
  Diarrhoea-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.17 | 0.04 | 0.08
  Diarrhoea-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Diarrhoea-non-SAE, R, Mild | 0.00 | 0.00 | 0.33 | 0.00 | 0.00 | 0.33
  Dyspepsia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Dyspnoea-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Ear Pain-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Exostosis-non-SAE, NR,Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Eye Infection Viral-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Eye Irritation-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Eye Oedema-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Fatigue-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Flatulence-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Flatulence-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Folliculitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Gastroenteritis Viral-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Headache-non-SAE, NR, Mild | 0.20 | 0.17 | 0.17 | 0.08 | 0.00 | 0.17
  Headache-non-SAE, R, Mild | 0.00 | 0.16 | 0.00 | 0.00 | 0.00 | 0.16
  Infection-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.04 | 0.10
  Influenza-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Infusion Site Haematoma-non-SAE, R, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Infusion Site Haemorrhage-non-SAE, R, Mild | 0.00 | 0.07 | 0.00 | 0.00 | 0.00 | 0.07
  Infusion Site Oedema-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Infusion Site Pain-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.00
  Infusion Site Pruritus-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Injection Site Haematoma-non-SAE, R, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Injection Site Pain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Joint Sprain-non-SAE, NR, Mild | 0.00 | 0.17 | 0.00 | 0.00 | 0.00 | 0.17
  Joint Swelling-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Joint Swelling-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Laryngitis Viral-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Limb Injury-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Lymphadenopathy-non-SAE, NR, Mild | 0.25 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Memory Impairment-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Migraine-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Migraine-non-SAE, R, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Muscle Strain-non-SAE, NR, Mild | 0.00 | 0.00 | 0.17 | 0.00 | 0.03 | 0.10
  Nasal Congestion-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Nasal Congestion-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Nasopharyngitis-non-SAE, NR, Mild | 0.25 | 0.08 | 0.00 | 0.00 | 0.04 | 0.04
  Nasopharyngitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.07 | 0.07
  Nausea-non-SAE, NR, Mild | 0.00 | 0.08 | 0.17 | 0.08 | 0.17 | 0.13
  Nausea-non-SAE, R, Mild | 0.00 | 0.08 | 0.17 | 0.00 | 0.04 | 0.08
  Nausea-non-SAE, R, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Oedema Peripheral-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Oral Herpes-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Oropharyngeal Pain-non-SAE, NR, Mild | 0.20 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Oropharyngeal Pain-non-SAE, NR, Moderate | 0.23 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Osteopenia-non-SAE, NR, Moderate | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Pain In Extremity-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Pharyngitis-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Pharyngitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Pneumonia-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Pneumonia Bacterial-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.17 | 0.00 | 0.00 | 0.17
  Pyrexia-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.04 | 0.06
  Rales-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Respir. Tract Infect. Viral-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Respir. Tract Infect Viral-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Sinusitis-non-SAE, NR, Mild | 0.00 | 0.00 | 0.00 | 0.00 | 0.04 | 0.04
  Sinusitis-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.17 | 0.08 | 0.00 | 0.17
  Sports Injury-non-SAE, NR, Mild | 0.00 | 0.08 | 0.00 | 0.00 | 0.00 | 0.08
  Upper Respir. Tract Infection-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.08 | 0.03 | 0.06
  Upper Respir. Tract Infect.-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Urinary Tract Infection-non-SAE, NR, Moderate | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Vestibulitis-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Viral Up. Respir Tract Infec-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08
  Vomiting-non-SAE, NR, Mild | 0.25 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Vulvovaginal Mycotic Infect.-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.00 | 0.03 | 0.03
  Wound-non-SAE, NR, Moderate | 0.00 | 0.00 | 0.00 | 0.08 | 0.00 | 0.08

35. Secondary Outcome: Percentage of Infusions Associated With ≥1 AE Related to the Study Drug
Time Frame: Throughout the study period (1 year and 9 months)
Population: All participants who received any study drug
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
Percentage of infusions
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 22.2 | 27.8 | 2.2
  Study Part 2 (SC) (N = 595, 469, 126) | 9.9 | 10.2 | 8.7
  Study Part 3a (SC) (N = 268, 206, 62) | 7.8 | 8.3 | 6.5
  Study Part 3b (SC) (N = 538, 418, 120) | 3.5 | 4.3 | 0.8
  Study Extension (SC) (N = 893, 664, 229) | 3.1 | 3.8 | 1.3
  Total SC (N = 2294, 1757, 537) | 5.5 | 6.1 | 3.5

36. Secondary Outcome: Percentage of Infusions Associated With ≥1 AEs That Begin During Infusion or Within 72 Hours of Completion of Infusion
Time Frame: During Infusion or Within 72 Hours of Completion of Infusions
Population: All participants who received any study drug
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
Percentage of infusions
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 30.9 | 35.8 | 13.3
  Study Part 2 (SC) (N = 595, 469, 126) | 15.0 | 15.8 | 11.9
  Study Part 3a (SC) (N = 268, 206, 62) | 11.6 | 12.6 | 8.1
  Study Part 3b (SC) (N = 538, 418, 120) | 8.7 | 8.9 | 8.3
  Study Extension (SC) (N = 893, 664, 229) | 9.4 | 10.5 | 6.1
  Total SC (N = 2294, 1757, 537) | 10.9 | 11.8 | 8.2

37. Secondary Outcome: Percentage of Infusions Associated With ≥1 AE Excluding Infections That Begin During Infusion or Within 72 Hours of Completion of Infusion.
Time Frame: During Infusion or Within 72 Hours of Completion of Infusions
Population: All participants who received any study drug
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
Percentage of infusions
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 28.5 | 32.7 | 13.3
  Study Part 2 (SC) (N = 595, 469, 126) | 11.8 | 12.2 | 10.3
  Study Part 3a (SC) (N = 268, 206, 62) | 10.1 | 11.2 | 6.5
  Study Part 3b (SC) (N = 538, 418, 120) | 7.2 | 7.2 | 7.5
  Study Extension (SC) (N = 893, 664, 229) | 7.3 | 8.1 | 4.8
  Total SC (N = 2294, 1757, 537) | 8.8 | 9.3 | 6.9

38. Secondary Outcome: Percentage of Infusions Associated With ≥1 Systemic AE Excluding Infections That Begin During Infusion or Within 72 Hours of Completion of Infusion.
Time Frame: During Infusion or Within 72 Hours of Completion of Infusions
Population: All participants who received any study drug
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
Percentage of infusions
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 28.0 | 32.1 | 13.3
  Study Part 2 (SC) (N = 595, 469, 126) | 7.6 | 7.7 | 7.1
  Study Part 3a (SC) (N = 268, 206, 62) | 7.8 | 8.3 | 6.5
  Study Part 3b (SC) (N = 538, 418, 120) | 6.1 | 5.7 | 7.5
  Study Extension (SC) (N = 893, 664, 229) | 6.3 | 6.9 | 4.4
  Total SC (N = 2294, 1757, 537) | 6.8 | 7.0 | 6.0

39. Primary Outcome: Percentage of Participants With Prior Experience With Subcutaneous Administration of Immunoglobulins (SESC) Who Had Any Infusion for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped
Description: as for outcome 19
Time Frame: Throughout study (1 year and 9 months)
Population: SESC data set (all participants with prior experience with subcutaneous administration of immunoglobulins who received any study drug)
Measure: Number; unit: Percentage of Participants
Arm/Group | Infusion Rate Change - For Any Reason | Infusion Rate Change - For Tolerability/AE
Number analyzed (Participants) | 11 | 11
Percentage of Participants
  Study Part 1 (IV) (n= 11) | 0.0 | 0.00
  Study Part 2 (SC) (n= 11) | 18.2 | 0.00
  Study Part 3A (SC) (n=10) | 0.00 | 0.00
  Study Part 3B (SC) (n=10) | 0.00 | 0.00
  Study Extension (SC) (n= 9) | 11.1 | 0.00
  Study Part 2, 3A, 3B, Study Extension (n= 11) | 18.2 | 0.00

40. Primary Outcome: Percentage of Infusions in FSDS for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped
Description: Ability to tolerate IGIV, 10% administered IV or SC. Measured as the percentage of infusions for which the infusion rate was reduced at any infusion and/or the infusion was interrupted or stopped for (i) any reason and (ii) for tolerability concerns or AEs
Time Frame: Throughout study (1 year and 9 months)
Population: Full safety data set (all participants who received any study drug)
Measure: Number (95% Confidence Interval); unit: Percentage of Infusions
Units Other Than Participants: Infusions
Groups:
- Infusion Rate Change (Percentage) - For Any Reason: Infusion Rate Reduced and/or Infusion Interrupted or Stopped. Percentage of Infusions with a change in the infusion rate.
- Infusion Rate Change - For Tolerability/AE: Infusion Rate Reduced and/or Infusion Interrupted or Stopped
Arm/Group | Infusion Rate Change (Percentage) - For Any Reason | Infusion Rate Change - For Tolerability/AE
Number analyzed (Participants) | 49 | 49
Number analyzed (Infusions) | 2501 | 2501
Percentage of Infusions
  Study Part 1 (IV) (n= 207 Infusions) | 6.7 [3.6 to 11.3] | 6.2 [3.2 to 10.5]
  Study Part 2 (SC) (n= 595 Infusions) | 4.2 [2.7 to 6.2] | 0.5 [0.1 to 1.3]
  Study Part 3A (SC) (n=268 Infusions) | 3.1 [1.4 to 5.8] | 0.4 [0.0 to 1.7]
  Study Part 3B (SC) (n=538 Infusions) | 1.1 [0.4 to 2.3] | 0.2 [0.0 to 0.8]
  Study Extension (SC) (n= 893 Infusions) | 0.6 [0.2 to 1.2] | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Parts 2, 3A, 3B, & Extension (n= 2,294 Infusions) | 1.9 [1.4 to 2.5] | 0.2 [0.1 to 0.5]

41. Primary Outcome: Percentage of Infusions in SNSC for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped
Description: as for outcome 40
Time Frame: Throughout study (1 year and 9 months)
Population: SNSC data set (all participants naïve to SC administration of immunoglobulins who received any study drug)
Measure: Number (95% Confidence Interval); unit: Percentage of Infusions
Units Other Than Participants: Infusions
Arm/Group | Infusion Rate Change (Percentage) - For Any Reason | Infusion Rate Change - For Tolerability/AE
Number analyzed (Participants) | 38 | 38
Number analyzed (Infusions) | 1919 | 1919
Percentage of Infusions
  Study Part 1 (IV) (n= 162 Infusions) | 8.7 [4.7 to 14.8] | 8.0 [4.2 to 13.8]
  Study Part 2 (SC) (n= 469 Infusions) | 4.5 [2.8 to 6.8] | 0.6 [0.2 to 1.7]
  Study Part 3A (SC) (n=206 Infusions) | 4.0 [1.8 to 7.7] | 0.5 [0.0 to 2.2]
  Study Part 3B (SC) (n=418 Infusions) | 1.5 [0.6 to 3.0] | 0.2 [0.0 to 1.1]
  Study Extension (SC) (n= 664 Infusions) | 0.6 [0.2 to 1.4] | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Parts 2, 3A, 3B, & Extension (n= 1,757 Infusions) | 2.2 [1.6 to 3.0] | 0.3 [0.1 to 0.6]

42. Primary Outcome: Percentage of Infusions in SESC for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped
Description: as for outcome 40
Time Frame: Throughout study (1 year and 9 months)
Population: as for outcome 39
Measure: Number (95% Confidence Interval); unit: Percentage of Infusions
Units Other Than Participants: Infusions
Arm/Group | Infusion Rate Change (Percentage) - For Any Reason | Infusion Rate Change - For Tolerability/AE
Number analyzed (Participants) | 11 | 11
Number analyzed (Infusions) | 582 | 582
Percentage of Infusions
  Study Part 1 (IV) (n= 45 Infusions) | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval. | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Study Part 2 (SC) (n= 126 Infusions) | 3.3 [1.0 to 7.8] | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Study Part 3A (SC) (n=62 Infusions) | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval. | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Study Part 3B (SC) (n=120 Infusions) | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval. | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Study Extension (SC) (n= 229 Infusions) | 0.4 [0.0 to 1.9] | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.
  Parts 2, 3A, 3B, & Extension (n= 537 Infusions) | 0.9 [0.3 to 2.0] | 0.0 [NA to NA] — There were no infusion rate changes; therefore there is no confidence interval.

43. Secondary Outcome: Percentage of Infusions Associated With ≥1 Local AE Excluding Infections That Begin During Infusion or Within 72 Hours of Completion of Infusion.
Time Frame: During Infusion or Within 72 Hours of Completion of Infusions
Population: All participants who received any study drug
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | FSDS | SNSC | SESC
Number analyzed (Participants) | 49 | 38 | 11
Number analyzed (Infusions) | 2501 | 1919 | 582
Percentage of infusions
  Study Part 1 (IV) (Units Analyzed N= 207, 162, 45) | 1.0 | 1.2 | 0.0
  Study Part 2 (SC) (N = 595, 469, 126) | 4.9 | 5.1 | 4.0
  Study Part 3a (SC) (N = 268, 206, 62) | 2.2 | 2.9 | 0.0
  Study Part 3b (SC) (N = 538, 418, 120) | 1.5 | 1.9 | 0.0
  Study Extension (SC) (N = 893, 664, 229) | 1.1 | 1.4 | 0.4
  Total SC (N = 2294, 1757, 537) | 2.3 | 2.7 | 1.1

ADVERSE EVENTS:
Time Frame: Throughout the entire study period (1 year, 9 months)
Groups:
- IV Treatment Period: Study Part 1
- SC Treatment Period: Study Parts 2, 3a, 3b, and Extension
Arm/Group | IV Treatment Period | SC Treatment Period
Serious Adverse Events (participants affected / at risk) | 2/49 | 2/48
Other Adverse Events (participants affected / at risk) | 38/49 | 44/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Treatment Period (N=49) | SC Treatment Period (N=48)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Convulsion/seizure (Nervous system disorders) | 1 (1) | 0 (0)
Biliary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Treatment Period (N=49) | SC Treatment Period (N=47)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 4 (5)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (2) | 5 (12)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 3 (4)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 3 (4)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 5 (13)
NAUSEA (Gastrointestinal disorders) | 5 (6) | 8 (22)
VOMITING (Gastrointestinal disorders) | 7 (11) | 7 (12)
CHILLS (General disorders) | 7 (13) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 7 (11)
INFUSION SITE ERYTHEMA (General disorders) | 0 (0) | 3 (3)
INFUSION SITE HAEMATOMA (General disorders) | 0 (0) | 5 (15)
INFUSION SITE OEDEMA (General disorders) | 0 (0) | 3 (3)
INFUSION SITE PAIN (General disorders) | 1 (2) | 10 (22)
INFUSION SITE RASH (General disorders) | 0 (0) | 4 (4)
PYREXIA (General disorders) | 5 (8) | 14 (22)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 1 (1) | 3 (10)
HEART RATE INCREASED (Investigations) | 4 (5) | 3 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (9)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3)
HEADACHE (Nervous system disorders) | 17 (42) | 23 (42)
MIGRAINE (Nervous system disorders) | 1 (1) | 4 (5)
SINUS HEADACHE (Nervous system disorders) | 2 (3) | 3 (3)
INSOMNIA (Psychiatric disorders) | 1 (1) | 3 (3)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (9)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (8)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)